CLINICAL TRIAL: NCT03703102
Title: A Phase 2, Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of an Anti-OX40 Monoclonal Antibody (KHK4083) in Subjects With Moderate to Severe Atopic Dermatitis (AD)
Brief Title: Study of an Anti-OX40 Monoclonal Antibody (KHK4083) in Subjects With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4083-006
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
Keywords: AD; eczema; skin diseases; biologics
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Skin Diseases | interventions — KHK4083

STUDY DESIGN:
Intervention Model Description: subcutaneous administration
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Placebo Comparator): Subcutaneous administration of placebo
  Interventions: Drug: Placebo
- Arm B (Experimental): Subcutaneous administration of KHK4083 (dose level 1, dosing regimen 2)
  Interventions: Drug: KHK4083
- Arm C (Experimental): Subcutaneous administration of KHK4083 (dose level 2, dosing regimen 1)
  Interventions: Drug: KHK4083
- Arm D (Experimental): Subcutaneous administration of KHK4083 (dose level 3, dosing regimen 1)
  Interventions: Drug: KHK4083
- Arm E (Experimental): Subcutaneous administration of KHK4083 (dose level 3, dosing regimen 2)
  Interventions: Drug: KHK4083

INTERVENTIONS:
Drug: KHK4083 — Anti-OX40 Monoclonal Antibody KHK4083
  Arms: Arm B; Arm C; Arm D; Arm E
Drug: Placebo — Matching placebo
  Arms: Arm A

SUMMARY:
A Phase 2, multicenter, randomized, placebo-controlled, double-blind, parallel-group study for subjects with moderate to severe AD whose disease cannot be adequately controlled with topical medications or for whom topical treatment is medically inadvisable.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent to participate in the study;
* Chronic AD, according to American Academy of Dermatology Consensus Criteria or the local diagnostic criteria, that has been present for at least 1 year before screening;
* EASI score ≥16 at screening and baseline;
* IGA score ≥3 (moderate) at both screening and baseline;
* BSA ≥10% at both screening and baseline;
* Documented recent history (within 1 year prior to screening visit) of inadequate response to treatment with topical medications or for whom topical treatments are otherwise medically inadvisable (e.g., because of important side effects or safety risks).

Exclusion Criteria:

* Current or past history of clinically significant illness(es) deemed by the Investigator to be likely to affect the study conduct and assessments. Examples include, but are not limited to, clinically significant cardiovascular (e.g., New York Heart Association [NYHA] Class III or IV), uncontrolled diabetes (HbA1c ≥9%), liver (e.g., Child-Pugh class B or C), renal, respiratory, hematologic, central nervous system, psychiatric, or autoimmune diseases/disorders;
* Any of the following laboratory abnormalities at screening:

  * Serum creatinine: >1.5 mg/dL
  * AST or ALT: ≥2.5 times the upper limit of normal (ULN)
  * Neutrophil count: <1.5×10³/μL
  * Other laboratory abnormalities that may affect the completion or evaluation of the study, as judged by the Investigator;
* Active malignancies, or onset or a history of treatment of malignancies within 5 years prior to informed consent (except curatively treated in situ cervical carcinoma, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehsanollah Esfandiari, MD, PhD, Study Director — Kyowa Kirin Pharmaceutical International Ltd.
Locations (58):
- United States (13):
  - Kyowa Investigational Site US-19, Huntington Beach, California
  - Kyowa Investigational Site US-17, Irvine, California
  - Kyowa Investigational Site US-09, Los Angeles, California
  - Kyowa Investigational Site US-05, Santa Ana, California
  - Kyowa Investigational Site US-10, Aurora, Colorado
  - Kyowa Investigational Site US-14, Clearwater, Florida
  - Kyowa Investigational Site US-04, Boston, Massachusetts
  - Kyowa Investigational Site US-01, New York, New York
  - Kyowa Investigational Site US-20, Charlotte, North Carolina
  - Kyowa Investigational Site US-11, Cleveland, Ohio
  - Kyowa Investigational Site US-08, Portland, Oregon
  - Kyowa Investigational Site US-02, Dallas, Texas
  - Kyowa Investigational Site US-07, Galveston, Texas
- Canada (6):
  - Kyowa Investigational Site CA-02, Markham, Ontario
  - Kyowa Investigational Site CA-03, Richmond Hill, Ontario
  - Kyowa Investigational Site CA-08, Richmond Hill, Ontario
  - Kyowa Investigational Site CA-07, Québec, Quebec
  - Kyowa Investigational Site CA-09, Québec, Quebec
  - Kyowa Investigational Site CA-04, Sherbrooke, Quebec
- Germany (8):
  - Kyowa Investigational Site GE-13, Aachen
  - Kyowa Investigational Site GE-07, Berlin
  - Kyowa Investigational Site GE-14, Berlin
  - Kyowa Investigational Site GE-08, Darmstadt
  - Kyowa Investigational Site GE-05, Frankfurt am Main
  - Kyowa Investigational Site GE-02, Hamburg
  - Kyowa Investigational Site GE-11, Hanover
  - Kyowa Investigational Site GE-01, Langenau
- Japan (31):
  - Kyowa Investigational Site JP-17, Aichi
  - Kyowa Investigational Site JP-27, Aichi
  - Kyowa Investigational Site JP-24, Chiba
  - Kyowa Investigational Site JP-08, Fukuoka
  - Kyowa Investigational Site JP-09, Fukuoka
  - Kyowa Investigational Site JP-12, Fukuoka
  - Kyowa Investigational Site JP-19, Fukuoka
  - Kyowa Investigational Site JP-26, Fukuoka
  - Kyowa Investigational Site JP-14, Gifu
  - Kyowa Investigational Site JP-01, Hokkaido
  - Kyowa Investigational Site JP-02, Hokkaido
  - Kyowa Investigational Site JP-04, Hokkaido
  - Kyowa Investigational Site JP-29, Hokkaido
  - Kyowa Investigational Site JP-31, Ibaraki
  - Kyowa Investigational Site JP-10, Kagoshima
  - Kyowa Investigational Site JP-11, Kagoshima
  - Kyowa Investigational Site JP-05, Kanagawa
  - Kyowa Investigational Site JP-06, Kanagawa
  - Kyowa Investigational Site JP-21, Kanagawa
  - Kyowa Investigational Site JP-18, Mie
  - Kyowa Investigational Site JP-20, Miyagi
  - Kyowa Investigational Site JP-28, Morioka
  - Kyowa Investigational Site JP-25, Shimane
  - Kyowa Investigational Site JP-15, Tochigi
  - Kyowa Investigational Site JP-03, Tokyo
  - Kyowa Investigational Site JP-07, Tokyo
  - Kyowa Investigational Site JP-13, Tokyo
  - Kyowa Investigational Site JP-16, Tokyo
  - Kyowa Investigational Site JP-22, Tokyo
  - Kyowa Investigational Site JP-23, Tokyo
  - Kyowa Investigational Site JP-30, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gooderham M, Guttman-Yassky E, Igawa K, Kabashima K, Esfandiari E, Rylands AJ, Williams A, Nixon A, Dent JE, Simpson E. Rocatinlimab Improves Patient-Reported Outcomes in Adults with Moderate-to-Severe Atopic Dermatitis: Results from a Double-Blind Placebo-Controlled Phase 2b Study. Dermatol Ther (Heidelb). 2024 Dec;14(12):3351-3366. doi: 10.1007/s13555-024-01303-z. Epub 2024 Nov 12. PMID 39532780
- [Derived] Guttman-Yassky E, Simpson EL, Reich K, Kabashima K, Igawa K, Suzuki T, Mano H, Matsui T, Esfandiari E, Furue M. An anti-OX40 antibody to treat moderate-to-severe atopic dermatitis: a multicentre, double-blind, placebo-controlled phase 2b study. Lancet. 2023 Jan 21;401(10372):204-214. doi: 10.1016/S0140-6736(22)02037-2. Epub 2022 Dec 9. PMID 36509097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The screening period began in September 2018. A total of 61 sites in four countries (Canada, Germany, Japan, and the United States) screened 351 patients and enrolled 274. The screening period closed in September 2019.
Pre-assignment Details: In Treatment Period A, randomized subjects received either study drug or placebo for 18 weeks. In Treatment Period B, the patients randomized to the placebo arm received study drug for 18 weeks. There was no treatment change for patients randomized to study drug arms.
  One subject who was randomized to the 600 mg Q4W group did not receive any study drug due to consent withdrawal before the start of the treatment. They are not included in baseline or any of the analysis sets.
Groups:
- KHK4083 150 mg SC Q4W: Subjects in this arm received 150 mg of KHK4083 at Weeks 0 (Day 1), 4, 8, 12, 16, 20, 24, 28, and 32.
  To maintain the blind, they received placebo at Weeks 2, 6, 10, 14, 18, 22, 26, 30, and 34.
- KHK4083 600 mg SC Q4W: Subjects in this arm received 600 mg of KHK4083 at Weeks 0 (Day 1), 4, 8, 12, 16, 20, 24, 28, and 32.
  To maintain the blind, they received placebo at Weeks 2, 6, 10, 14, 18, 22, 26, 30, and 34.
- KHK4083 300 mg SC Q2W: Subjects in this arm received 300 mg of KHK4083 at Weeks 0 (Day 1), 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, and 34.
- KHK4083 600 mg SC Q2W: Subjects in this arm received 600 mg of KHK4083 at Weeks 0 (Day 1), 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, and 34.
- Placebo/KHK4083 600 mg: Subjects in this arm received placebo at Weeks 0 (Day 1), 2, 4, 6, 8, 10, 12, 14, and 16, and received KHK4083 600 mg at Weeks 18 (Day 127), 20, 22, 24, 26, 28, 30, 32, and 34.
Period: Overall Study
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Started | 54 | 53 | 55 | 54 | 57
Completed Treatment Period A | 42 | 41 | 42 | 46 | 34
Completed Treatment Period B | 33 | 39 | 37 | 38 | 26
Completed | 32 | 38 | 33 | 37 | 24
Not Completed | 22 | 15 | 22 | 17 | 33
Not completed — Adverse Event | 4 | 3 | 7 | 3 | 13
Not completed — Lack of Efficacy | 4 | 0 | 1 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 2
Not completed — Physician Decision | 2 | 2 | 2 | 2 | 4
Not completed — Withdrawal by Subject | 7 | 5 | 5 | 5 | 9
Not completed — Ineligibility | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 4 | 4 | 3 | 0 | 0
Not completed — Non-Compliance with Study Drug | 1 | 1 | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Population: One subject who was randomized to the 600 mg Q4W group did not receive any study treatment due to consent withdrawal before the start of the treatment. They are not included in baseline or any of the analysis sets.
Groups:
- Total: Total of all reporting groups
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg | Total
Number analyzed (Participants) | 54 | 53 | 55 | 54 | 57 | 273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 51 | 51 | 49 | 52 | 255
  >=65 years | 2 | 2 | 4 | 5 | 5 | 18
Age, Continuous [Mean (Full Range); unit: years] | 37.4 [19 to 67] | 38.9 [18 to 70] | 37.5 [18 to 77] | 37.3 [18 to 89] | 38.7 [18 to 69] | 38.0 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 24 | 24 | 26 | 113
  Male | 37 | 31 | 31 | 30 | 31 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 1 | 1 | 7
  Not Hispanic or Latino | 51 | 51 | 54 | 53 | 54 | 263
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 36 | 32 | 37 | 33 | 37 | 175
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 2 | 1 | 6 | 13
  White | 14 | 20 | 16 | 20 | 14 | 84
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 5 | 5 | 4 | 7 | 25
  United States | 11 | 10 | 11 | 11 | 13 | 56
  Japan | 32 | 30 | 33 | 32 | 32 | 159
  Germany | 7 | 8 | 6 | 7 | 5 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 16 in Eczema Area and Severity Index (EASI) Score
Description: In the EASI assessment, the severity of 4 elements of eczema (erythema, induration/papulation, excoriation, and lichenification) at each of 4 body regions (head and neck, trunk, upper extremities, and lower extremities) will be assessed on a scale of 0 to 3 (0 = None , 1 = Mild, 2 = Moderate, 3 = Severe). Half scores (1.5 and 2.5) are allowed, with the exception of 0.5. Any signs must be at least 1 (mild) in severity. In addition, the extent of eczema at each of the 4 body regions will be assessed on a scale of 0 to 6 (0 = 0%, 1 = 1% to 9%, 2 = 10% to 29%, 3 = 30% to 49%, 4 = 50% to 69%, 5 = 70% to 89%, 6 = 90% to 100%). Scores calculated according to the expression "total score of 4 elements of eczema × area score of eczema" will be multiplied by 0.1 for head and neck, 0.2 for upper extremities, 0.3 for trunk, and 0.4 for lower extremities. The 4 region scores obtained will then be summed up (maximum score: 72) as EASI score.
Time Frame: Baseline to Week 16
Population: Full analysis set: One subject in the 600 mg Q4W group was excluded from all analysis sets as the subject was not exposed to IP. Two subjects in the 150 mg Q4W group, 1 subject in the 600 mg Q4W group, and 3 subjects in the 300 mg Q2W group were excluded from the full analysis set. Those 6 subjects had no evaluable EASI score after the start of IP administration until Week 16.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change | -48.33 [-62.62 to -34.04] | -49.72 [-62.47 to -35.17] | -61.07 [-75.19 to -46.96] | -57.35 [-71.27 to -43.43] | -15.01 [-28.60 to -1.43]
Statistical Analysis 1: Comparison: KHK4083 150 mg SC Q4W vs Placebo/KHK4083 600 mg; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: KHK4083 600 mg SC Q4W vs Placebo/KHK4083 600 mg; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: KHK4083 300 mg SC Q2W vs Placebo/KHK4083 600 mg; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: KHK4083 600 mg SC Q2W vs Placebo/KHK4083 600 mg; Test type: Superiority; p < 0.001, ANCOVA

2. Secondary Outcome: Achievement of 50%, 75%, or 90% Reduction From Baseline in Eczema Area and Severity Index (EASI) Score (EASI-50, EASI-75, or EASI-90) at Week 16
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
Participants
  Achieved EASI-50 at Week 16 | 30 | 31 | 36 | 35 | 17
  achieved EASI-75 at Week 16 | 23 | 21 | 28 | 21 | 6
  achieved EASI-90 at Week 16 | 10 | 6 | 19 | 10 | 2

3. Secondary Outcome: Change From Baseline to Week 16 in Eczema Area and Severity Index (EASI) Score
Description: as for outcome 1
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale | -22.5 (14.7) | -20.7 (14.3) | -23.3 (9.0) | -19.9 (11.8) | -9.8 (13.0)

4. Secondary Outcome: Change From Baseline to Week 16 in SCORing Atopic Dermatitis (SCORAD) Score
Description: In the SCORAD assessment, the extent of AD will be calculated as the sum of the percentage of each defined body area, with a maximum score of 100% (assigned as "A" in the overall SCORAD calculation). The severity of 6 specific symptoms of AD will be assessed using the following scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe, with a maximum score of 18 (assigned as "B" in the overall SCORAD calculation). Itch and sleeplessness will be assessed by subjects on a visual analogue scale (VAS), where 0 is no itch (or sleeplessness) and 10 is the worst imaginable itch (or sleeplessness), with a maximum score of 20 (assigned as "C" in the overall SCORAD calculation). The SCORAD score is calculated as A/5 + 7B/2 + C. The maximum possible SCORAD score is 103; higher scores indicate poorer or more severe condition.
Time Frame: Baseline to Week 16
Population: Full analysis set: One subject in the 600 mg Q4W group was excluded from all analysis sets as the subject was not exposed to IP. Two subjects in the 150 mg Q4W group, 1 subject in the 600 mg Q4W group, and 3 subjects in the 300 mg Q2W group were excluded from the full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale | -23.71 [-30.72 to -16.69] | -23.86 [-30.92 to -16.81] | -30.44 [-37.27 to -23.61] | -27.65 [-34.39 to -20.91] | -8.09 [-14.65 to -1.53]

5. Secondary Outcome: Percent Change From Baseline to Week 16 in SCORing Atopic Dermatitis (SCORAD) Score
Description: as for outcome 4
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change | -34.86 [-45.20 to -24.51] | -35.13 [-45.54 to -24.72] | -46.69 [-56.77 to -36.61] | -40.76 [-50.70 to -30.81] | -11.90 [-21.59 to -2.22]

6. Secondary Outcome: Achievement of an Investigator's Global Assessment (IGA) Score of 0 or 1 and a Reduction From Baseline of ≥2 Points at Week 16
Description: In the IGA, the Investigator will evaluate the overall skin symptoms of subjects at each visit on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
Participants | 10 | 8 | 16 | 10 | 1

7. Secondary Outcome: Change From Baseline to Week 16 in Percent Body Surface Area of Involvement of AD (BSA)
Description: The Investigator will calculate the percentage (%) of the total body surface area affected by AD.
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of total BSA involvement
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of total BSA involvement | -22.86 [-30.30 to -15.42] | -21.48 [-29.07 to -13.89] | -27.92 [-35.30 to -20.54] | -25.04 [-32.33 to -17.76] | -7.87 [-14.96 to -0.77]

8. Secondary Outcome: Change From Baseline to Week 16 in Pruritus Numerical Rating Scale (NRS) Score
Description: The worst degree of itch experienced during 24 hours before the time point will be assessed on a Numerical Rating Scale. The degree of itch will be scored on an 11-point scale, with 0 being "no itch" and 10 being the "worst itch imaginable."
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale | -2.04 [-2.90 to -1.18] | -3.02 [-3.90 to -2.15] | -3.60 [-4.44 to -2.75] | -2.81 [-3.64 to -1.97] | -1.31 [-2.12 to -0.49]

9. Secondary Outcome: Percent Change From Baseline to Week 16 in Pruritus Numerical Rating Scale (NRS) Score
Description: as for outcome 8
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change | -25.57 [-39.48 to -11.66] | -34.38 [-48.56 to -20.21] | -47.99 [-61.71 to -34.26] | -36.83 [-50.41 to -23.25] | -6.18 [-6.18 to 7.01]

10. Secondary Outcome: Change From Baseline to Week 16 in Sleep Disturbance Numerical Rating Scale (NRS) Score
Description: Daily sleep disturbance in the last 24 hours before the relevant time point will be assessed on a Numerical Rating Scale. Subjects will score the degree of their sleep disturbance on an 11-point scale ranging from 'no sleep loss' (0) to 'I cannot sleep at all' (10).
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale | -1.09 [-2.01 to -0.18] | -1.93 [-2.86 to -1.00] | -2.59 [-3.48 to -1.69] | -2.00 [-2.90 to -1.11] | -0.01 [-0.87 to 0.86]

11. Secondary Outcome: Percent Change From Baseline to Week 16 in Sleep Disturbance Numerical Rating Scale (NRS) Score
Description: as for outcome 10
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change | -8.19 [-44.32 to 27.95] | -7.02 [-44.96 to 30.93] | -41.58 [-78.30 to -4.86] | -33.17 [-69.08 to 2.74] | -46.54 [-100.55 to -8.89]

12. Secondary Outcome: Change From Baseline to Week 16 in Dermatology Life Quality Index (DLQI)
Description: DLQI consists of 6 subscales (symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment), which are scored from 0 to 3 on the basis of 10 questions. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more QoL is impaired.
Time Frame: Baseline to Week 16
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale | -2.59 [-4.73 to -0.44] | -4.66 [-6.89 to -2.43] | -6.28 [-8.38 to -4.18] | -4.93 [-7.01 to -2.84] | 0.19 [-1.88 to 2.27]

13. Secondary Outcome: EASI Score at Each Time Point
Description: as for outcome 1
Time Frame: 56 Weeks
Population: The overall number of participants analyzed is the number of subjects in the full analysis set. The number of participants analyzed per row is the number of patients who had values at the specified time points.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- KHK4083 150 mg SC Q4W: Subjects in this arm received 150 mg of KHK4083 at Weeks 0 (Day 1), 4, 8, 12, 16, 20, 24, 28, and 32.
  To maintain the blind, they received placebo at Weeks 2, 6, 10, 14, 18, 22, 26, 30, and 34.
  Weeks 40-56 visits are off-treatment.
- KHK4083 600 mg SC Q4W: Subjects in this arm received 600 mg of KHK4083 at Weeks 0 (Day 1), 4, 8, 12, 16, 20, 24, 28, and 32.
  To maintain the blind, they received placebo at Weeks 2, 6, 10, 14, 18, 22, 26, 30, and 34.
  Weeks 40-56 visits are off-treatment.
- KHK4083 300 mg SC Q2W: Subjects in this arm received 300 mg of KHK4083 at Weeks 0 (Day 1), 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, and 34.
  Weeks 40-56 visits are off-treatment.
- KHK4083 600 mg SC Q2W: Subjects in this arm received 600 mg of KHK4083 at Weeks 0 (Day 1), 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, and 34.
  Weeks 40-56 visits are off-treatment.
- Placebo/KHK4083 600 mg: Subjects in this arm received placebo at Weeks 0 (Day 1), 2, 4, 6, 8, 10, 12, 14, and 16, and received KHK4083 600 mg at Weeks 18 (Day 127), 20, 22, 24, 26, 28, 30, 32, and 34.
  Weeks 40-56 visits are off-treatment.
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale
  EASI Score at Baseline | 33.2 [16 to 63] | 32.5 [16 to 69] | 31.6 [16 to 64] | 31.1 [16 to 60] | 29.2 [16 to 68]
  EASI Score at Week 1: number analyzed (Participants) | 50 | 51 | 50 | 54 | 54
  EASI Score at Week 1 | 33.0 [10 to 65] | 29.5 [6 to 58] | 28.6 [6 to 69] | 29.4 [2 to 57] | 28.5 [6 to 62]
  EASI Score at Week 2: number analyzed (Participants) | 46 | 50 | 48 | 53 | 50
  EASI Score at Week 2 | 31.7 [5 to 67] | 27.6 [6 to 60] | 25.6 [2 to 66] | 27.2 [0 to 58] | 28.1 [5 to 71]
  EASI Score at Week 4: number analyzed (Participants) | 46 | 49 | 46 | 52 | 44
  EASI Score at Week 4 | 27.3 [0 to 71] | 26.3 [5 to 56] | 22.4 [2 to 49] | 23.4 [1 to 68] | 28.8 [2 to 71]
  EASI Score at Week 6: number analyzed (Participants) | 42 | 48 | 42 | 51 | 41
  EASI Score at Week 6 | 24.7 [0 to 66] | 21.6 [0 to 57] | 17.6 [0 to 52] | 19.6 [0 to 52] | 27.9 [2 to 71]
  EASI Score at Week 8: number analyzed (Participants) | 42 | 45 | 42 | 50 | 40
  EASI Score at Week 8 | 20.3 [0 to 63] | 17.6 [0 to 55] | 15.2 [1 to 50] | 17.3 [0 to 51] | 25.8 [3 to 67]
  EASI Score at Week 10: number analyzed (Participants) | 43 | 44 | 43 | 48 | 39
  EASI Score at Week 10 | 16.5 [0 to 72] | 15.8 [0 to 65] | 12.9 [0 to 47] | 16.1 [0 to 46] | 25.5 [2 to 72]
  EASI Score at Week 12: number analyzed (Participants) | 43 | 45 | 42 | 48 | 36
  EASI Score at Week 12 | 14.7 [0 to 72] | 13.9 [0 to 53] | 10.5 [0 to 47] | 14.9 [1 to 45] | 23.6 [1 to 72]
  EASI Score at Week 14: number analyzed (Participants) | 42 | 42 | 42 | 48 | 34
  EASI Score at Week 14 | 12.6 [0 to 62] | 12.6 [0 to 55] | 9.8 [0 to 45] | 12.1 [0 to 44] | 22.7 [1 to 71]
  EASI Score at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  EASI Score at Week 15 | 10.8 [0 to 59] | 12.6 [0 to 50] | 9.0 [0 to 48] | 11.6 [0 to 37] | 20.6 [0 to 72]
  EASI Score at Week 16: number analyzed (Participants) | 41 | 44 | 43 | 47 | 36
  EASI Score at Week 16 | 10.8 [0 to 62] | 11.8 [0 to 48] | 8.0 [0 to 40] | 11.1 [0 to 41] | 20.4 [0 to 72]
  EASI Score at Week 18: number analyzed (Participants) | 41 | 43 | 40 | 46 | 33
  EASI Score at Week 18 | 10.5 [0 to 60] | 11.0 [0 to 41] | 8.7 [0 to 39] | 10.6 [0 to 60] | 22.2 [0 to 72]
  EASI Score at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  EASI Score at Week 20 | 10.0 [0 to 72] | 9.5 [0 to 39] | 7.2 [0 to 32] | 8.1 [0 to 38] | 20.8 [0 to 62]
  EASI Score at Week 22: number analyzed (Participants) | 39 | 40 | 41 | 44 | 31
  EASI Score at Week 22 | 8.9 [0 to 72] | 7.5 [0 to 37] | 6.5 [0 to 38] | 6.0 [0 to 36] | 16.6 [0 to 60]
  EASI Score at Week 24: number analyzed (Participants) | 40 | 40 | 41 | 42 | 30
  EASI Score at Week 24 | 9.4 [0 to 72] | 7.4 [0 to 37] | 5.0 [0 to 37] | 6.2 [0 to 46] | 15.9 [0 to 53]
  EASI Score at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 26
  EASI Score at Week 26 | 8.2 [0 to 72] | 6.8 [0 to 35] | 4.3 [0 to 36] | 5.8 [0 to 46] | 10.8 [0 to 48]
  EASI Score at Week 28: number analyzed (Participants) | 36 | 38 | 38 | 40 | 26
  EASI Score at Week 28 | 7.7 [0 to 72] | 6.8 [0 to 29] | 4.7 [0 to 37] | 4.8 [0 to 28] | 9.8 [0 to 46]
  EASI Score at Week 30: number analyzed (Participants) | 34 | 37 | 38 | 40 | 25
  EASI Score at Week 30 | 6.5 [0 to 51] | 6.1 [0 to 26] | 4.1 [0 to 50] | 3.8 [0 to 24] | 8.4 [0 to 38]
  EASI Score at Week 32: number analyzed (Participants) | 33 | 38 | 37 | 40 | 23
  EASI Score at Week 32 | 6.4 [0 to 64] | 5.2 [0 to 25] | 2.9 [0 to 20] | 3.3 [0 to 18] | 6.3 [0 to 27]
  EASI Score at Week 34: number analyzed (Participants) | 33 | 38 | 35 | 37 | 23
  EASI Score at Week 34 | 5.9 [0 to 67] | 5.8 [0 to 27] | 2.6 [0 to 19] | 3.4 [0 to 29] | 5.7 [0 to 30]
  EASI Score at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 37 | 25
  EASI Score at Week 36 | 5.6 [0 to 62] | 4.8 [0 to 26] | 2.1 [0 to 16] | 3.5 [0 to 17] | 6.3 [0 to 42]
  EASI Score at Week 40: number analyzed (Participants) | 26 | 34 | 30 | 30 | 22
  EASI Score at Week 40 | 4.1 [0 to 25] | 3.8 [0 to 21] | 2.7 [0 to 30] | 3.1 [0 to 13] | 5.5 [0 to 30]
  EASI Score at Week 44: number analyzed (Participants) | 24 | 34 | 29 | 30 | 19
  EASI Score at Week 44 | 3.5 [0 to 30] | 5.8 [0 to 72] | 1.5 [0 to 9] | 3.1 [0 to 12] | 2.8 [0 to 17]
  EASI Score at Week 48: number analyzed (Participants) | 22 | 32 | 28 | 26 | 17
  EASI Score at Week 48 | 6.5 [0 to 33] | 3.0 [0 to 20] | 1.6 [0 to 7] | 2.5 [0 to 12] | 3.2 [0 to 19]
  EASI Score at Week 52: number analyzed (Participants) | 18 | 33 | 23 | 24 | 17
  EASI Score at Week 52 | 3.1 [0 to 12] | 2.9 [0 to 20] | 2.2 [0 to 19] | 2.3 [0 to 10] | 2.6 [0 to 9]
  EASI Score at Week 56: number analyzed (Participants) | 19 | 28 | 18 | 20 | 16
  EASI Score at Week 56 | 4.2 [0 to 22] | 4.7 [0 to 32] | 2.4 [0 to 18] | 2.8 [0 to 14] | 3.2 [0 to 11]

14. Secondary Outcome: Percent Change From Baseline in EASI Score at Each Time Point
Description: as for outcome 1
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change
  EASI Score % Change at Week 1: number analyzed (Participants) | 50 | 51 | 50 | 54 | 54
  EASI Score % Change at Week 1 | -2.5 [-55 to 48] | -9.5 [-68 to 31] | -8.5 [-72 to 100] | -7.0 [-89 to 96] | -2.9 [-63 to 114]
  EASI Score % Change at Week 2: number analyzed (Participants) | 46 | 50 | 48 | 53 | 50
  EASI Score % Change at Week 2 | -6.7 [-71 to 71] | -14.3 [-75 to 31] | -18.4 [-88 to 128] | -15.6 [-100 to 79] | -2.6 [-72 to 154]
  EASI Score % Change at Week 4: number analyzed (Participants) | 46 | 49 | 46 | 52 | 44
  EASI Score % Change at Week 4 | -19.6 [-100 to 78] | -19.4 [-74 to 42] | -26.4 [-92 to 167] | -24.6 [-96 to 57] | -8.5 [-89 to 58]
  EASI Score % Change at Week 6: number analyzed (Participants) | 42 | 48 | 42 | 51 | 41
  EASI Score % Change at Week 6 | -28.8 [-100 to 48] | -32.5 [-100 to 54] | -43.4 [-100 to 94] | -35.8 [-100 to 70] | -11.1 [-89 to 76]
  EASI Score % Change at Week 8: number analyzed (Participants) | 42 | 45 | 42 | 50 | 40
  EASI Score % Change at Week 8 | -40.3 [-100 to 118] | -45.5 [-100 to 29] | -52.2 [-97 to 37] | -42.1 [-100 to 50] | -19.2 [-83 to 150]
  EASI Score % Change at Week 10: number analyzed (Participants) | 43 | 44 | 43 | 48 | 39
  EASI Score % Change at Week 10 | -51.5 [-100 to 45] | -51.9 [-100 to 86] | -60.4 [-100 to 25] | -48.2 [-100 to 50] | -21.1 [-91 to 66]
  EASI Score % Change at Week 12: number analyzed (Participants) | 43 | 45 | 42 | 48 | 36
  EASI Score % Change at Week 12 | -56.7 [-100 to 24] | -58.4 [-100 to 9] | -68.3 [-100 to 26] | -50.9 [-96 to 12] | -29.5 [-95 to 61]
  EASI Score % Change at Week 14: number analyzed (Participants) | 42 | 42 | 42 | 48 | 34
  EASI Score % Change at Week 14 | -62.5 [-100 to 7] | -62.1 [-100 to 12] | -71.1 [-100 to 36] | -61.5 [-100 to 0] | -32.1 [-95 to 30]
  EASI Score % Change at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  EASI Score % Change at Week 15 | -67.1 [-100 to 2] | -62.2 [-100 to 6] | -74.1 [-100 to -9] | -62.6 [-100 to 19] | -35.3 [-100 to 81]
  EASI Score % Change at Week 16: number analyzed (Participants) | 41 | 44 | 43 | 47 | 36
  EASI Score % Change at Week 16 | -67.0 [-100 to 18] | -63.2 [-100 to 6] | -77.2 [-100 to -20] | -63.6 [-100 to 52] | -37.4 [-100 to 81]
  EASI Score % Change at Week 18: number analyzed (Participants) | 41 | 43 | 40 | 46 | 33
  EASI Score % Change at Week 18 | -67.1 [-100 to 10] | -66.1 [-100 to -6] | -75.5 [-100 to -13] | -63.9 [-100 to 233] | -32.6 [-100 to 81]
  EASI Score % Change at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  EASI Score % Change at Week 20 | -69.7 [-100 to 24] | -70.6 [-100 to 0] | -79.0 [-100 to -12] | -74.4 [-100 to 11] | -37.9 [-100 to 95]
  EASI Score % Change at Week 22: number analyzed (Participants) | 39 | 40 | 41 | 44 | 31
  EASI Score % Change at Week 22 | -74.3 [-100 to 24] | -75.6 [-100 to -5] | -80.8 [-100 to -12] | -79.4 [-100 to 33] | -49.3 [-100 to 95]
  EASI Score % Change at Week 24: number analyzed (Participants) | 40 | 40 | 41 | 42 | 30
  EASI Score % Change at Week 24 | -71.7 [-100 to 24] | -75.5 [-100 to -5] | -85.3 [-100 to 9] | -80.4 [-100 to 15] | -49.7 [-100 to 105]
  EASI Score % Change at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 26
  EASI Score % Change at Week 26 | -75.3 [-100 to 24] | -78.2 [-100 to -23] | -86.3 [-100 to -18] | -81.0 [-100 to 15] | -70.1 [-100 to 20]
  EASI Score % Change at Week 28: number analyzed (Participants) | 36 | 38 | 38 | 40 | 26
  EASI Score % Change at Week 28 | -78.7 [-100 to 24] | -77.5 [-100 to -20] | -84.8 [-100 to 32] | -83.9 [-100 to -7] | -70.6 [-100 to 15]
  EASI Score % Change at Week 30: number analyzed (Participants) | 34 | 37 | 38 | 40 | 25
  EASI Score % Change at Week 30 | -80.8 [-100 to -12] | -81.1 [-100 to -31] | -87.3 [-100 to 11] | -86.5 [-100 to -14] | -74.5 [-100 to -6]
  EASI Score % Change at Week 32: number analyzed (Participants) | 33 | 38 | 37 | 40 | 23
  EASI Score % Change at Week 32 | -82.5 [-100 to 10] | -82.7 [-100 to -31] | -90.5 [-100 to -56] | -87.9 [-100 to -36] | -82.4 [-100 to -44]
  EASI Score % Change at Week 34: number analyzed (Participants) | 33 | 38 | 35 | 37 | 23
  EASI Score % Change at Week 34 | -83.6 [-100 to 16] | -80.5 [-100 to -23] | -91.3 [-100 to -52] | -87.1 [-100 to 4] | -81.8 [-100 to -18]
  EASI Score % Change at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 37 | 25
  EASI Score % Change at Week 36 | -84.5 [-100 to 7] | -83.5 [-100 to -24] | -93.0 [-100 to -62] | -87.2 [-100 to -39] | -82.2 [-100 to 5]
  EASI Score % Change at Week 40: number analyzed (Participants) | 26 | 34 | 30 | 30 | 22
  EASI Score % Change at Week 40 | -88.0 [-100 to -36] | -86.9 [-100 to -52] | -91.7 [-100 to -33] | -88.4 [-100 to -54] | -82.3 [-100 to 0]
  EASI Score % Change at Week 44: number analyzed (Participants) | 24 | 34 | 29 | 30 | 19
  EASI Score % Change at Week 44 | -89.1 [-100 to -14] | -81.7 [-100 to 106] | -94.8 [-100 to -82] | -88.5 [-100 to -41] | -86.7 [-100 to 0]
  EASI Score % Change at Week 48: number analyzed (Participants) | 22 | 32 | 28 | 26 | 17
  EASI Score % Change at Week 48 | -84.5 [-100 to -11] | -90.8 [-100 to -56] | -94.3 [-100 to -78] | -91.6 [-100 to -57] | -85.0 [-100 to 12]
  EASI Score % Change at Week 52: number analyzed (Participants) | 18 | 33 | 23 | 24 | 17
  EASI Score % Change at Week 52 | -90.4 [-100 to -42] | -92.2 [-100 to -56] | -93.2 [-100 to -66] | -92.4 [-100 to -58] | -90.2 [-100 to -63]
  EASI Score % Change at Week 56: number analyzed (Participants) | 19 | 28 | 18 | 20 | 16
  EASI Score % Change at Week 56 | -87.4 [-100 to -32] | -88.3 [-100 to -35] | -90.3 [-100 to -36] | -90.4 [-100 to -57] | -88.3 [-100 to -50]

15. Secondary Outcome: Achievement of EASI-50, EASI-75, or EASI-90 at Each Time Point
Description: In the EASI assessment, the severity of 4 elements of eczema (erythema, induration/papulation, excoriation, and lichenification) at each of 4 body regions (head and neck, trunk, upper extremities, and lower extremities) will be assessed on a scale of 0 to 3 (0 = None , 1 = Mild, 2 = Moderate, 3 = Severe). Half scores (1.5 and 2.5) are allowed, with the exception of 0.5. Any signs must be at least 1 (mild) in severity. In addition, the extent of eczema at each of the 4 body regions will be assessed on a scale of 0 to 6 (0 = 0%, 1 = 1% to 9%, 2 = 10% to 29%, 3 = 30% to 49%, 4 = 50% to 69%, 5 = 70% to 89%, 6 = 90% to 100%).
Time Frame: 56 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
Participants
  Achievement of EASI-50 at Week 1 | 1 | 2 | 7 | 3 | 1
  Achievement of EASI-50 at Week 2 | 5 | 7 | 11 | 8 | 3
  Achievement of EASI-50 at Week 4 | 10 | 9 | 14 | 11 | 2
  Achievement of EASI-50 at Week 6 | 12 | 17 | 22 | 20 | 5
  Achievement of EASI-50 at Week 8 | 18 | 21 | 29 | 24 | 10
  Achievement of EASI-50 at Week 10 | 26 | 29 | 32 | 26 | 10
  Achievement of EASI-50 at Week 12 | 28 | 31 | 34 | 27 | 13
  Achievement of EASI-50 at Week 14 | 31 | 31 | 33 | 34 | 12
  Achievement of EASI-50 at Week 15 | 30 | 30 | 33 | 31 | 15
  Achievement of EASI-50 at Week 16 | 30 | 31 | 36 | 35 | 17
  Achievement of EASI-50 at Week 18 | 32 | 32 | 34 | 36 | 16
  Achievement of EASI-50 at Week 20 | 33 | 32 | 36 | 39 | 17
  Achievement of EASI-50 at Week 22 | 32 | 34 | 36 | 41 | 19
  Achievement of EASI-50 at Week 24 | 32 | 34 | 39 | 40 | 19
  Achievement of EASI-50 at Week 26 | 31 | 31 | 35 | 39 | 21
  Achievement of EASI-50 at Week 28 | 30 | 33 | 34 | 38 | 21
  Achievement of EASI-50 at Week 30 | 30 | 35 | 36 | 39 | 21
  Achievement of EASI-50 at Week 32 | 30 | 35 | 37 | 38 | 21
  Achievement of EASI-50 at Week 34 | 31 | 36 | 35 | 35 | 20
  Achievement of EASI-50 at Week 36 | 31 | 34 | 36 | 36 | 23
  Achievement of EASI-50 at Week 40 | 24 | 34 | 29 | 30 | 20
  Achievement of EASI-50 at Week 44 | 23 | 31 | 29 | 29 | 18
  Achievement of EASI-50 at Week 48 | 19 | 32 | 28 | 26 | 16
  Achievement of EASI-50 at Week 52 | 17 | 33 | 23 | 24 | 17
  Achievement of EASI-50 at Week 56 | 18 | 25 | 17 | 20 | 16
  Achievement of EASI-75 at Week 1 | 0 | 0 | 0 | 1 | 0
  Achievement of EASI-75 at Week 2 | 0 | 1 | 3 | 3 | 0
  Achievement of EASI-75 at Week 4 | 6 | 0 | 6 | 7 | 1
  Achievement of EASI-75 at Week 6 | 5 | 5 | 12 | 8 | 2
  Achievement of EASI-75 at Week 8 | 11 | 7 | 10 | 11 | 3
  Achievement of EASI-75 at Week 10 | 11 | 11 | 17 | 13 | 5
  Achievement of EASI-75 at Week 12 | 13 | 14 | 24 | 16 | 4
  Achievement of EASI-75 at Week 14 | 17 | 17 | 25 | 17 | 5
  Achievement of EASI-75 at Week 15 | 19 | 18 | 25 | 18 | 7
  Achievement of EASI-75 at Week 16 | 23 | 21 | 28 | 21 | 6
  Achievement of EASI-75 at Week 18 | 22 | 21 | 26 | 27 | 8
  Achievement of EASI-75 at Week 20 | 24 | 21 | 26 | 27 | 8
  Achievement of EASI-75 at Week 22 | 27 | 29 | 30 | 30 | 11
  Achievement of EASI-75 at Week 24 | 25 | 28 | 34 | 29 | 11
  Achievement of EASI-75 at Week 26 | 25 | 29 | 34 | 33 | 17
  Achievement of EASI-75 at Week 28 | 26 | 26 | 33 | 32 | 17
  Achievement of EASI-75 at Week 30 | 24 | 26 | 32 | 32 | 18
  Achievement of EASI-75 at Week 32 | 23 | 29 | 31 | 35 | 19
  Achievement of EASI-75 at Week 34 | 23 | 27 | 30 | 31 | 19
  Achievement of EASI-75 at Week 36 | 27 | 30 | 33 | 31 | 20
  Achievement of EASI-75 at Week 40 | 23 | 28 | 27 | 26 | 17
  Achievement of EASI-75 at Week 44 | 21 | 27 | 29 | 25 | 17
  Achievement of EASI-75 at Week 48 | 19 | 30 | 28 | 24 | 15
  Achievement of EASI-75 at Week 52 | 16 | 30 | 22 | 22 | 14
  Achievement of EASI-75 at Week 56 | 15 | 24 | 16 | 17 | 14
  Achievement of EASI-90 at Week 1 | 0 | 0 | 0 | 0 | 0
  Achievement of EASI-90 at Week 2 | 0 | 0 | 0 | 2 | 0
  Achievement of EASI-90 at Week 4 | 2 | 0 | 1 | 2 | 0
  Achievement of EASI-90 at Week 6 | 2 | 1 | 3 | 2 | 0
  Achievement of EASI-90 at Week 8 | 4 | 3 | 7 | 4 | 0
  Achievement of EASI-90 at Week 10 | 7 | 3 | 8 | 5 | 1
  Achievement of EASI-90 at Week 12 | 9 | 4 | 10 | 5 | 26
  Achievement of EASI-90 at Week 14 | 6 | 6 | 16 | 8 | 2
  Achievement of EASI-90 at Week 15 | 11 | 6 | 17 | 8 | 3
  Achievement of EASI-90 at Week 16 | 10 | 6 | 19 | 10 | 2
  Achievement of EASI-90 at Week 18 | 9 | 11 | 15 | 13 | 3
  Achievement of EASI-90 at Week 20 | 14 | 14 | 17 | 14 | 3
  Achievement of EASI-90 at Week 22 | 16 | 15 | 20 | 17 | 5
  Achievement of EASI-90 at Week 24 | 14 | 14 | 26 | 16 | 6
  Achievement of EASI-90 at Week 26 | 14 | 16 | 26 | 20 | 6
  Achievement of EASI-90 at Week 28 | 15 | 14 | 25 | 17 | 5
  Achievement of EASI-90 at Week 30 | 14 | 18 | 25 | 24 | 8
  Achievement of EASI-90 at Week 32 | 16 | 17 | 27 | 25 | 11
  Achievement of EASI-90 at Week 34 | 19 | 15 | 27 | 24 | 11
  Achievement of EASI-90 at Week 36 | 18 | 19 | 28 | 21 | 13
  Achievement of EASI-90 at Week 40 | 15 | 19 | 23 | 18 | 13
  Achievement of EASI-90 at Week 44 | 14 | 24 | 24 | 20 | 12
  Achievement of EASI-90 at Week 48 | 14 | 21 | 22 | 18 | 11
  Achievement of EASI-90 at Week 52 | 12 | 24 | 17 | 19 | 11
  Achievement of EASI-90 at Week 56 | 13 | 21 | 13 | 15 | 8

16. Secondary Outcome: SCORing Atopic Dermatitis (SCORAD) Score at Each Time Point
Description: as for outcome 4
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Median (Full Range); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale
  SCORAD Score at Baseline: number analyzed (Participants) | 51 | 52 | 52 | 54 | 57
  SCORAD Score at Baseline | 68.67 [42.0 to 96.3] | 69.80 [42.9 to 99.6] | 68.19 [42.1 to 96.4] | 68.79 [40.1 to 100.2] | 66.35 [38.7 to 97.8]
  SCORAD Score at Week 1: number analyzed (Participants) | 50 | 51 | 50 | 54 | 54
  SCORAD Score at Week 1 | 68.40 [29.0 to 97.8] | 66.53 [34.5 to 95.3] | 63.06 [28.5 to 97.7] | 64.99 [22.5 to 99.6] | 62.83 [26.2 to 94.1]
  SCORAD Score at Week 2: number analyzed (Participants) | 46 | 50 | 48 | 52 | 50
  SCORAD Score at Week 2 | 64.56 [21.3 to 98.7] | 62.75 [27.1 to 96.8] | 61.03 [30.8 to 97.1] | 62.52 [1.8 to 97.1] | 65.31 [28.1 to 103.7]
  SCORAD Score at Week 4: number analyzed (Participants) | 46 | 49 | 45 | 52 | 44
  SCORAD Score at Week 4 | 60.87 [10.5 to 98.7] | 59.84 [24.6 to 99.9] | 54.01 [18.7 to 95.3] | 57.01 [16.4 to 99.0] | 65.20 [24.8 to 98.2]
  SCORAD Score at Week 6: number analyzed (Participants) | 42 | 48 | 42 | 51 | 41
  SCORAD Score at Week 6 | 56.59 [0.9 to 101.5] | 52.39 [10.0 to 88.7] | 46.32 [8.2 to 82.9] | 51.34 [11.9 to 93.6] | 62.07 [19.9 to 99.2]
  SCORAD Score at Week 8: number analyzed (Participants) | 42 | 44 | 42 | 50 | 40
  SCORAD Score at Week 8 | 48.46 [1.0 to 101.4] | 48.16 [7.5 to 87.6] | 45.05 [16.8 to 84.5] | 48.29 [10.2 to 94.4] | 59.11 [26.0 to 103.4]
  SCORAD Score at Week 10: number analyzed (Participants) | 43 | 44 | 43 | 48 | 39
  SCORAD Score at Week 10 | 42.42 [0.6 to 100.7] | 45.15 [7.4 to 85.7] | 39.13 [0.6 to 75.8] | 45.50 [9.4 to 90.1] | 58.85 [20.3 to 103.1]
  SCORAD Score at Week 12: number analyzed (Participants) | 43 | 45 | 42 | 48 | 36
  SCORAD Score at Week 12 | 41.07 [1.3 to 102.5] | 41.98 [8.0 to 84.9] | 33.82 [4.0 to 68.0] | 43.68 [9.7 to 89.4] | 57.15 [15.3 to 102.9]
  SCORAD Score at Week 14: number analyzed (Participants) | 42 | 42 | 42 | 48 | 34
  SCORAD Score at Week 14 | 39.51 [1.3 to 101.6] | 39.75 [11.7 to 88.9] | 31.69 [3.8 to 67.6] | 39.41 [1.0 to 88.1] | 54.68 [14.1 to 96.4]
  SCORAD Score at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  SCORAD Score at Week 15 | 35.79 [0.5 to 93.7] | 38.88 [2.3 to 81.9] | 30.03 [0.5 to 76.9] | 37.46 [0.9 to 69.3] | 51.66 [16.7 to 96.8]
  SCORAD Score at Week 16: number analyzed (Participants) | 40 | 44 | 43 | 47 | 36
  SCORAD Score at Week 16 | 34.70 [0.8 to 97.8] | 37.82 [2.0 to 77.8] | 28.31 [3.5 to 70.1] | 35.76 [1.1 to 72.4] | 51.80 [16.3 to 97.0]
  SCORAD Score at Week 18: number analyzed (Participants) | 40 | 43 | 39 | 46 | 33
  SCORAD Score at Week 18 | 36.44 [0.4 to 97.8] | 36.01 [1.4 to 71.3] | 30.14 [0.3 to 64.5] | 34.80 [6.2 to 83.8] | 51.99 [19.6 to 97.6]
  SCORAD Score at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  SCORAD Score at Week 20 | 33.88 [0.3 to 100.3] | 33.86 [1.3 to 63.8] | 27.59 [0.2 to 66.4] | 31.35 [0.2 to 74.2] | 48.17 [13.0 to 90.6]
  SCORAD Score at Week 22: number analyzed (Participants) | 39 | 40 | 41 | 44 | 31
  SCORAD Score at Week 22 | 31.69 [0.3 to 98.9] | 30.13 [0.1 to 59.4] | 25.14 [0.2 to 57.5] | 28.21 [0.2 to 64.0] | 45.07 [0.6 to 88.8]
  SCORAD Score at Week 24: number analyzed (Participants) | 40 | 40 | 41 | 41 | 30
  SCORAD Score at Week 24 | 32.41 [0.4 to 98.5] | 29.06 [0.1 to 57.0] | 21.05 [0.2 to 59.3] | 29.93 [0.2 to 93.8] | 43.55 [8.0 to 90.8]
  SCORAD Score at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 26
  SCORAD Score at Week 26 | 29.48 [0.3 to 101.9] | 27.54 [0.3 to 56.5] | 20.12 [0.0 to 66.5] | 28.31 [0.2 to 93.0] | 35.59 [4.3 to 80.6]
  SCORAD Score at Week 28: number analyzed (Participants) | 36 | 38 | 38 | 40 | 26
  SCORAD Score at Week 28 | 29.21 [0.2 to 102.7] | 27.50 [1.7 to 55.7] | 20.23 [0.1 to 68.0] | 27.05 [0.2 to 68.2] | 32.88 [11.3 to 74.1]
  SCORAD Score at Week 30: number analyzed (Participants) | 34 | 37 | 38 | 40 | 25
  SCORAD Score at Week 30 | 25.75 [0.2 to 79.2] | 25.40 [0.3 to 50.7] | 18.05 [0.2 to 59.2] | 23.79 [0.2 to 58.6] | 33.63 [10.9 to 76.1]
  SCORAD Score at Week 32: number analyzed (Participants) | 33 | 38 | 36 | 40 | 23
  SCORAD Score at Week 32 | 25.09 [0.2 to 102.2] | 25.02 [0.2 to 48.3] | 16.29 [0.0 to 48.0] | 22.05 [0.1 to 46.4] | 29.23 [8.8 to 69.8]
  SCORAD Score at Week 34: number analyzed (Participants) | 33 | 37 | 35 | 37 | 23
  SCORAD Score at Week 34 | 24.63 [0.2 to 102.4] | 25.78 [0.4 to 49.2] | 15.65 [0.0 to 40.9] | 22.13 [0.5 to 58.5] | 27.55 [6.6 to 76.6]
  SCORAD Score at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 36 | 25
  SCORAD Score at Week 36 | 23.82 [0.2 to 93.8] | 24.13 [0.2 to 56.7] | 15.46 [0.0 to 39.2] | 23.78 [0.4 to 51.8] | 26.86 [10.3 to 73.6]
  SCORAD Score at Week 40: number analyzed (Participants) | 26 | 34 | 30 | 30 | 22
  SCORAD Score at Week 40 | 20.98 [0.1 to 54.3] | 21.49 [0.4 to 46.6] | 15.56 [0.1 to 59.3] | 24.14 [1.1 to 48.0] | 22.27 [0.3 to 59.8]
  SCORAD Score at Week 44: number analyzed (Participants) | 24 | 33 | 29 | 30 | 19
  SCORAD Score at Week 44 | 18.33 [0.2 to 66.5] | 21.86 [0.4 to 92.8] | 11.64 [0.1 to 34.8] | 20.08 [0.1 to 52.0] | 17.72 [0.4 to 61.8]
  SCORAD Score at Week 48: number analyzed (Participants) | 21 | 31 | 28 | 26 | 16
  SCORAD Score at Week 48 | 25.83 [0.1 to 67.3] | 17.78 [0.1 to 45.0] | 11.90 [0.0 to 40.2] | 18.54 [0.1 to 39.1] | 17.54 [0.5 to 62.2]
  SCORAD Score at Week 52: number analyzed (Participants) | 18 | 32 | 23 | 24 | 17
  SCORAD Score at Week 52 | 19.96 [0.3 to 42.5] | 16.60 [0.0 to 62.6] | 15.02 [0.0 to 66.3] | 20.46 [0.1 to 47.4] | 15.21 [0.2 to 37.3]
  SCORAD Score at Week 56: number analyzed (Participants) | 19 | 28 | 17 | 20 | 16
  SCORAD Score at Week 56 | 20.65 [0.5 to 60.3] | 18.50 [0.2 to 76.0] | 11.92 [0.0 to 61.1] | 19.27 [0.1 to 43.3] | 16.91 [0.4 to 34.3]

17. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Each Time Point
Description: as for outcome 4
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change
  SCORAD Score % Change at Week 1: number analyzed (Participants) | 49 | 51 | 50 | 54 | 54
  SCORAD Score % Change at Week 1 | -1.28 [-35.6 to 50.0] | -4.08 [-42.9 to 19.7] | -7.03 [-58.3 to 36.1] | -5.75 [-50.6 to 27.7] | -4.54 [-38.8 to 20.3]
  SCORAD Score % Change at Week 2: number analyzed (Participants) | 45 | 50 | 48 | 52 | 50
  SCORAD Score % Change at Week 2 | -7.37 [-52.7 to 31.7] | -9.14 [-61.8 to 35.2] | -9.05 [-53.4 to 18.2] | -10.37 [-95.9 to 32.8] | -0.47 [-34.8 to 45.0]
  SCORAD Score % Change at Week 4: number analyzed (Participants) | 45 | 49 | 45 | 52 | 44
  SCORAD Score % Change at Week 4 | -13.51 [-76.4 to 41.0] | -12.97 [-54.0 to 36.2] | -19.60 [-72.2 to 39.5] | -15.77 [-79.7 to 40.0] | -1.98 [-42.1 to 41.9]
  SCORAD Score % Change at Week 6: number analyzed (Participants) | 41 | 48 | 42 | 51 | 41
  SCORAD Score % Change at Week 6 | -19.34 [-98.0 to 45.0] | -23.76 [-86.1 to 20.3] | -30.52 [-73.0 to 15.5] | -29.34 [-85.3 to 28.5] | -12.34 [-53.5 to 74.8]
  SCORAD Score % Change at Week 8: number analyzed (Participants) | 41 | 44 | 42 | 50 | 40
  SCORAD Score % Change at Week 8 | -31.63 [-97.8 to 44.9] | -29.29 [-89.6 to 28.1] | -32.82 [-73.0 to 15.5] | -29.34 [-85.3 to 28.5] | -12.34 [-53.5 to 74.8]
  SCORAD Score % Change at Week 10: number analyzed (Participants) | 42 | 44 | 43 | 48 | 39
  SCORAD Score % Change at Week 10 | -39.55 [-98.7 to 13.7] | -34.22 [-89.7 to 28.1] | -42.53 [-99.1 to -0.5] | -34.32 [-86.5 to 4.6] | -13.14 [-63.7 to 21.3]
  SCORAD Score % Change at Week 12: number analyzed (Participants) | 42 | 45 | 42 | 48 | 36
  SCORAD Score % Change at Week 12 | -41.68 [-97.1 to 11.0] | -38.06 [-88.9 to 17.1] | -49.86 [-95.1 to 0.9] | -35.85 [-86.1 to 7.0] | -15.56 [-72.6 to 13.8]
  SCORAD Score % Change at Week 14: number analyzed (Participants) | 41 | 42 | 42 | 48 | 34
  SCORAD Score % Change at Week 14 | -44.39 [-97.3 to 7.9] | -41.69 [-83.8 to 18.2] | -53.03 [-95.4 to 7.4] | -42.09 [-98.7 to 16.3] | -19.05 [-74.8 to 24.7]
  SCORAD Score % Change at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  SCORAD Score % Change at Week 15 | -48.84 [-98.9 to -0.8] | -42.54 [-96.2 to 11.5] | -55.95 [-99.3 to -7.4] | -44.36 [-98.8 to 8.5] | -23.19 [-70.1 to 40.4]
  SCORAD Score % Change at Week 16: number analyzed (Participants) | 40 | 44 | 43 | 47 | 36
  SCORAD Score % Change at Week 16 | -50.07 [-98.5 to 3.5] | -43.47 [-96.7 to 18.9] | -58.24 [-95.8 to -13.9] | -47.00 [-98.5 to 12.1] | -23.26 [-71.7 to 42.9]
  SCORAD Score % Change at Week 18: number analyzed (Participants) | 40 | 43 | 39 | 46 | 33
  SCORAD Score % Change at Week 18 | -47.48 [-99.2 to 7.1] | -46.42 [-97.7 to 20.8] | -56.06 [-99.5 to -5.0] | -48.32 [-91.8 to 79.0] | -21.87 [-80.0 to 69.0]
  SCORAD Score % Change at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  SCORAD Score % Change at Week 20 | -51.55 [-99.4 to 10.0] | -49.39 [-97.9 to 17.8] | -58.91 [-99.7 to -2.8] | -54.95 [-99.7 to 9.6] | -27.64 [-85.7 to 76.6]
  SCORAD Score % Change at Week 22: number analyzed (Participants) | 39 | 40 | 41 | 44 | 31
  SCORAD Score % Change at Week 22 | -54.91 [-99.4 to 13.3] | -55.22 [-99.8 to 26.9] | -62.02 [-99.7 to -10.4] | -58.18 [-99.7 to -0.9] | -32.18 [-99.4 to 73.1]
  SCORAD Score % Change at Week 24: number analyzed (Participants) | 40 | 40 | 41 | 41 | 30
  SCORAD Score % Change at Week 24 | -53.96 [-99.2 to 13.6] | -56.56 [-99.8 to 2.3] | -68.56 [-99.7 to -3.4] | -56.63 [-99.7 to 5.7] | -34.10 [-86.3 to 77.0]
  SCORAD Score % Change at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 26
  SCORAD Score % Change at Week 26 | -58.23 [-99.4 to 7.8] | -59.24 [-99.5 to -13.5] | -68.82 [-100.0 to -3.5] | -58.19 [-99.7 to 4.8] | -47.60 [-92.6 to 18.8]
  SCORAD Score % Change at Week 28: number analyzed (Participants) | 36 | 38 | 38 | 40 | 26
  SCORAD Score % Change at Week 28 | -58.86 [-99.6 to 8.7] | -58.76 [-97.2 to -12.0] | -68.19 [-99.8 to -1.3] | -59.99 [-99.7 to 8.9] | -50.43 [-81.0 to 5.9]
  SCORAD Score % Change at Week 30: number analyzed (Participants) | 34 | 37 | 38 | 40 | 25
  SCORAD Score % Change at Week 30 | -63.35 [-99.6 to -8.1] | -62.81 [-99.5 to -30.2] | -72.05 [-99.7 to -7.8] | -64.57 [-99.7 to -20.2] | -49.89 [-76.6 to 14.6]
  SCORAD Score % Change at Week 32: number analyzed (Participants) | 33 | 38 | 36 | 40 | 23
  SCORAD Score % Change at Week 32 | -64.78 [-99.6 to 8.1] | -62.61 [-99.7 to -24.5] | -74.40 [-100.0 to -14.9] | -67.09 [-99.9 to -27.5] | -57.60 [-87.5 to -14.6]
  SCORAD Score % Change at Week 34: number analyzed (Participants) | 33 | 37 | 35 | 37 | 23
  SCORAD Score % Change at Week 34 | -64.71 [-99.6 to 8.4] | -61.29 [-99.3 to 7.5] | -75.43 [-100.0 to -31.5] | -66.43 [-99.3 to -10.7] | -59.75 [-92.3 to 8.7]
  SCORAD Score % Change at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 36 | 25
  SCORAD Score % Change at Week 36 | -65.54 [-99.7 to -0.7] | -63.75 [-99.6 to 29.5] | -75.38 [-100.0 to -22.5] | -64.60 [-99.5 to -22.9] | -60.63 [-87.3 to -1.8]
  SCORAD Score % Change at Week 40: number analyzed (Participants) | 26 | 34 | 30 | 30 | 22
  SCORAD Score % Change at Week 40 | -69.85 [-99.8 to -13.5] | -66.90 [-99.5 to 6.4] | -75.95 [-99.8 to -7.6] | -64.59 [-98.5 to -30.0] | -66.66 [-99.5 to -19.4]
  SCORAD Score % Change at Week 44: number analyzed (Participants) | 24 | 33 | 29 | 30 | 19
  SCORAD Score % Change at Week 44 | -74.31 [-99.6 to -3.5] | -67.86 [-99.5 to 39.3] | -80.96 [-99.9 to -31.2] | -70.81 [-99.8 to -18.2] | -71.50 [-99.4 to 3.2]
  SCORAD Score % Change at Week 48: number analyzed (Participants) | 21 | 31 | 28 | 26 | 16
  SCORAD Score % Change at Week 48 | -64.22 [-99.8 to -4.5] | -74.60 [-99.8 to -34.0] | -81.00 [-100.0 to -20.6] | -74.06 [-99.9 to -39.9] | -71.99 [-99.2 to 3.8]
  SCORAD Score % Change at Week 52: number analyzed (Participants) | 18 | 32 | 23 | 24 | 17
  SCORAD Score % Change at Week 52 | -70.53 [-99.4 to -23.1] | -76.82 [-100.0 to -16.8] | -77.96 [-100.0 to -12.0] | -71.47 [-99.9 to -38.1] | -76.93 [-99.6 to -39.9]
  SCORAD Score % Change at Week 56: number analyzed (Participants) | 19 | 28 | 17 | 20 | 16
  SCORAD Score % Change at Week 56 | -70.50 [-99.1 to -24.8] | -74.01 [-99.7 to 1.1] | -80.81 [-100.0 to -7.3] | -71.83 [-99.9 to -35.2] | -74.51 [-99.3 to -39.3]

18. Secondary Outcome: Achievement of an Investigator's Global Assessment (IGA) Score of 0 or 1 and a Reduction From Baseline of ≥2 Points at Each Time Point
Description: as for outcome 6
Time Frame: 56 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
Participants
  Achievement of IGA Score at Week 1 | 0 | 0 | 0 | 0 | 0
  Achievement of IGA Score at Week 2 | 0 | 0 | 1 | 1 | 0
  Achievement of IGA Score at Week 4 | 1 | 1 | 0 | 3 | 1
  Achievement of IGA Score at Week 6 | 2 | 2 | 1 | 2 | 0
  Achievement of IGA Score at Week 8 | 5 | 2 | 2 | 2 | 0
  Achievement of IGA Score at Week 10 | 6 | 4 | 6 | 2 | 1
  Achievement of IGA Score at Week 12 | 9 | 6 | 12 | 4 | 1
  Achievement of IGA Score at Week 14 | 8 | 5 | 11 | 4 | 2
  Achievement of IGA Score at Week 15 | 10 | 7 | 9 | 8 | 2
  Achievement of IGA Score at Week 16 | 10 | 8 | 16 | 10 | 1
  Achievement of IGA Score at Week 18 | 10 | 8 | 16 | 12 | 1
  Achievement of IGA Score at Week 20 | 13 | 9 | 15 | 14 | 3
  Achievement of IGA Score at Week 22 | 13 | 12 | 18 | 14 | 3
  Achievement of IGA Score at Week 24 | 14 | 10 | 20 | 12 | 3
  Achievement of IGA Score at Week 26 | 13 | 14 | 25 | 18 | 4
  Achievement of IGA Score at Week 28 | 11 | 12 | 23 | 14 | 3
  Achievement of IGA Score at Week 30 | 13 | 12 | 22 | 17 | 4
  Achievement of IGA Score at Week 32 | 14 | 13 | 24 | 23 | 5
  Achievement of IGA Score at Week 34 | 16 | 11 | 24 | 20 | 7
  Achievement of IGA Score at Week 36 | 18 | 14 | 27 | 19 | 8
  Achievement of IGA Score at Week 40 | 10 | 17 | 19 | 13 | 7
  Achievement of IGA Score at Week 44 | 12 | 16 | 25 | 16 | 11
  Achievement of IGA Score at Week 48 | 8 | 21 | 20 | 18 | 9
  Achievement of IGA Score at Week 52 | 10 | 19 | 18 | 15 | 10
  Achievement of IGA Score at Week 56 | 12 | 18 | 13 | 14 | 9

19. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) at Each Time Point
Description: The Investigator will calculate the percentage (%) of the total body surface area affected by AD.
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: percentage of total BSA involvement
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of total BSA involvement
  Change in % BSA at Week 1: number analyzed (Participants) | 50 | 51 | 50 | 54 | 54
  Change in % BSA at Week 1 | -0.5 [-25 to 17] | -1.4 [-25 to 23] | -0.4 [-35 to 40] | -0.1 [-23 to 23] | -1.2 [-35 to 45]
  Change in % BSA at Week 2: number analyzed (Participants) | 46 | 50 | 48 | 53 | 50
  Change in % BSA at Week 2 | -2.6 [-42 to 20] | -3.8 [-48 to 15] | -6.4 [-45 to 25] | -1.9 [-24 to 38] | 0.1 [-38 to 50]
  Change in % BSA at Week 4: number analyzed (Participants) | 46 | 49 | 46 | 52 | 44
  Change in % BSA at Week 4 | -6.7 [-60 to 35] | -4.0 [-48 to 39] | -10.7 [-63 to 25] | -5.6 [-49 to 23] | -2.2 [-27 to 20]
  Change in % BSA at Week 6: number analyzed (Participants) | 42 | 48 | 41 | 51 | 41
  Change in % BSA at Week 6 | -13.7 [-60 to 30] | -11.2 [-63 to 22] | -16.9 [-68 to 25] | -12.1 [-55 to 42] | -4.0 [-35 to 20]
  Change in % BSA at Week 8: number analyzed (Participants) | 42 | 45 | 42 | 50 | 40
  Change in % BSA at Week 8 | -18.6 [-70 to 32] | -19.3 [-76 to 6] | -21.4 [-73 to 25] | -17.2 [-55 to 25] | -4.4 [-33 to 40]
  Change in % BSA at Week 10: number analyzed (Participants) | 43 | 44 | 43 | 48 | 39
  Change in % BSA at Week 10 | -24.5 [-71 to 39] | -22.6 [-68 to 3] | -26.0 [-73 to 25] | -20.7 [-65 to 19] | -4.8 [-35 to 20]
  Change in % BSA at Week 12: number analyzed (Participants) | 43 | 45 | 41 | 48 | 36
  Change in % BSA at Week 12 | -27.4 [-75 to 39] | -26.4 [-73 to 5] | -31.1 [-77 to 25] | -22.2 [-72 to 22] | -4.9 [-35 to 20]
  Change in % BSA at Week 14: number analyzed (Participants) | 42 | 42 | 41 | 48 | 34
  Change in % BSA at Week 14 | -29.8 [-75 to 35] | -29.4 [-88 to 3] | -33.6 [-77 to 28] | -24.4 [-75 to 22] | -10.2 [-61 to 13]
  Change in % BSA at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  Change in % BSA at Week 15 | -31.9 [-75 to 24] | -29.3 [-79 to 2] | -35.1 [-81 to 15] | -25.6 [-75 to 32] | -12.2 [-61 to 20]
  Change in % BSA at Week 16: number analyzed (Participants) | 41 | 44 | 43 | 47 | 36
  Change in % BSA at Week 16 | -31.9 [-75 to 39] | -29.6 [-89 to 25] | -35.5 [-78 to 20] | -28.9 [-80 to 24] | -14.1 [-60 to 20]
  Change in % BSA at Week 18: number analyzed (Participants) | 41 | 43 | 40 | 46 | 33
  Change in % BSA at Week 18 | -34.6 [-80 to 39] | -32.7 [-89 to 0] | -35.5 [-75 to 5] | -29.6 [-86 to 39] | -13.1 [-60 to 30]
  Change in % BSA at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  Change in % BSA at Week 20 | -35.9 [-90 to 39] | -34.8 [-84 to 2] | -39.7 [-70 to 7] | -34.6 [-86 to 19] | -13.3 [-70 to 35]
  Change in % BSA at Week 22: number analyzed (Participants) | 39 | 40 | 41 | 44 | 31
  Change in % BSA at Week 22 | -39.3 [-94 to 39] | -38.3 [-84 to 0] | -40.6 [-77 to 11] | -38.3 [-80 to 21] | -18.5 [-95 to 35]
  Change in % BSA at Week 24: number analyzed (Participants) | 40 | 40 | 40 | 42 | 30
  Change in % BSA at Week 24 | -37.7 [-91 to 39] | -39.0 [-79 to 0] | -42.9 [-75 to 20] | -40.6 [-80 to 10] | -21.1 [-75 to 37]
  Change in % BSA at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 26
  Change in % BSA at Week 26 | -38.3 [-85 to 39] | -42.1 [-81 to -5] | -46.4 [-88 to -10] | -42.0 [-82 to 27] | -26.9 [-80 to 9]
  Change in % BSA at Week 28: number analyzed (Participants) | 36 | 38 | 37 | 40 | 25
  Change in % BSA at Week 28 | -41.2 [-90 to 34] | -43.1 [-83 to -5] | -45.8 [-87 to 3] | -42.8 [-78 to 37] | -29.6 [-70 to 7]
  Change in % BSA at Week 30: number analyzed (Participants) | 34 | 37 | 38 | 40 | 25
  Change in % BSA at Week 30 | -41.4 [-93 to 19] | -45.5 [-89 to -10] | -46.2 [-87 to -5] | -47.2 [-80 to -8] | -32.1 [-70 to 6]
  Change in % BSA at Week 32: number analyzed (Participants) | 33 | 38 | 37 | 40 | 23
  Change in % BSA at Week 32 | -44.0 [-90 to 39] | -46.5 [-89 to -7] | -48.3 [-85 to -15] | -48.2 [-84 to -3] | -39.6 [-80 to -9]
  Change in % BSA at Week 34: number analyzed (Participants) | 33 | 38 | 35 | 37 | 23
  Change in % BSA at Week 34 | -44.4 [-92 to 39] | -45.1 [-94 to -2] | -50.7 [-90 to -18] | -49.0 [-80 to -3] | -41.2 [-85 to -3]
  Change in % BSA at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 37 | 25
  Change in % BSA at Week 36 | -44.6 [-93 to 39] | -48.1 [-89 to 4] | -50.3 [-92 to -17] | -48.0 [-84 to -3] | -40.8 [-95 to 4]
  Change in % BSA at Week 40: number analyzed (Participants) | 26 | 33 | 30 | 30 | 21
  Change in % BSA at Week 40 | -49.0 [-95 to -5] | -50.6 [-87 to -4] | -51.6 [-92 to -18] | -51.1 [-82 to -4] | -46.6 [-99 to -1]
  Change in % BSA at Week 44: number analyzed (Participants) | 24 | 34 | 29 | 30 | 19
  Change in % BSA at Week 44 | -50.8 [-95 to -13] | -47.9 [-88 to 5] | -53.5 [-90 to -18] | -50.8 [-90 to 4] | -47.5 [-89 to -10]
  Change in % BSA at Week 48: number analyzed (Participants) | 22 | 32 | 28 | 26 | 17
  Change in % BSA at Week 48 | -46.6 [-87 to -12] | -52.7 [-89 to -13] | -53.9 [-90 to -18] | -53.7 [-90 to -24] | -46.2 [-90 to 0]
  Change in % BSA at Week 52: number analyzed (Participants) | 18 | 33 | 23 | 24 | 17
  Change in % BSA at Week 52 | -49.7 [-87 to -20] | -51.9 [-89 to -12] | -53.7 [-90 to -18] | -55.8 [-90 to -24] | -48.6 [-90 to -9]
  Change in % BSA at Week 56: number analyzed (Participants) | 19 | 28 | 18 | 20 | 16
  Change in % BSA at Week 56 | -45.6 [-80 to -10] | -47.2 [-89 to 3] | -53.8 [-90 to -18] | -58.6 [-90 to -27] | -45.9 [-85 to -6]

20. Secondary Outcome: Pruritus Numerical Rating Scale (NRS) Score at Each Time Point
Description: as for outcome 8
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale
  Pruritis NRS Score at Baseline | 7.7 [3 to 10] | 7.7 [2 to 10] | 7.3 [3 to 10] | 7.6 [1 to 10] | 7.2 [1 to 10]
  Pruritis NRS Score at Week 1: number analyzed (Participants) | 50 | 52 | 51 | 54 | 54
  Pruritis NRS Score at Week 1 | 7.3 [2 to 10] | 7.3 [2 to 10] | 6.8 [1 to 10] | 6.8 [1 to 10] | 6.9 [1 to 10]
  Pruritis NRS Score at Week 2: number analyzed (Participants) | 46 | 51 | 48 | 53 | 50
  Pruritis NRS Score at Week 2 | 6.8 [2 to 10] | 7.0 [2 to 10] | 6.3 [2 to 10] | 6.8 [1 to 10] | 7.1 [2 to 10]
  Pruritis NRS Score at Week 4: number analyzed (Participants) | 46 | 49 | 46 | 52 | 44
  Pruritis NRS Score at Week 4 | 6.4 [1 to 10] | 6.2 [1 to 10] | 5.7 [0 to 10] | 6.2 [1 to 10] | 7.1 [3 to 10]
  Pruritis NRS Score at Week 6: number analyzed (Participants) | 42 | 48 | 42 | 51 | 41
  Pruritis NRS Score at Week 6 | 6.0 [1 to 10] | 5.4 [0 to 10] | 4.7 [0 to 10] | 5.5 [0 to 10] | 6.5 [1 to 10]
  Pruritis NRS Score at Week 8: number analyzed (Participants) | 42 | 45 | 42 | 50 | 40
  Pruritis NRS Score at Week 8 | 5.4 [1 to 10] | 5.2 [0 to 10] | 4.4 [0 to 9] | 5.2 [1 to 10] | 6.0 [1 to 10]
  Pruritis NRS Score at Week 10: number analyzed (Participants) | 43 | 44 | 43 | 48 | 39
  Pruritis NRS Score at Week 10 | 4.9 [1 to 9] | 4.7 [0 to 10] | 4.0 [0 to 9] | 5.1 [1 to 10] | 5.8 [1 to 10]
  Pruritis NRS Score at Week 12: number analyzed (Participants) | 43 | 45 | 42 | 48 | 36
  Pruritis NRS Score at Week 12 | 4.8 [0 to 9] | 4.2 [0 to 10] | 3.6 [0 to 10] | 4.7 [1 to 10] | 5.8 [1 to 10]
  Pruritis NRS Score at Week 14: number analyzed (Participants) | 42 | 42 | 42 | 48 | 34
  Pruritis NRS Score at Week 14 | 4.5 [1 to 9] | 3.7 [0 to 10] | 3.3 [0 to 9] | 4.6 [1 to 10] | 5.9 [1 to 10]
  Pruritis NRS Score at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  Pruritis NRS Score at Week 15 | 4.4 [1 to 9] | 3.8 [0 to 10] | 2.9 [0 to 9] | 4.2 [1 to 9] | 5.3 [1 to 10]
  Pruritis NRS Score at Week 16: number analyzed (Participants) | 41 | 44 | 43 | 46 | 36
  Pruritis NRS Score at Week 16 | 4.6 [1 to 9] | 3.6 [0 to 10] | 2.8 [0 to 9] | 4.1 [0 to 9] | 5.2 [0 to 10]
  Pruritis NRS Score at Week 18: number analyzed (Participants) | 41 | 43 | 40 | 46 | 33
  Pruritis NRS Score at Week 18 | 4.2 [1 to 9] | 3.7 [0 to 10] | 3.3 [0 to 8] | 4.2 [0 to 10] | 5.2 [0 to 9]
  Pruritis NRS Score at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  Pruritis NRS Score at Week 20 | 4.0 [1 to 10] | 3.2 [0 to 10] | 2.9 [0 to 8] | 3.7 [0 to 10] | 4.8 [0 to 9]
  Pruritis NRS Score at Week 22: number analyzed (Participants) | 39 | 40 | 42 | 45 | 31
  Pruritis NRS Score at Week 22 | 4.0 [0 to 9] | 3.1 [0 to 10] | 2.3 [0 to 7] | 3.5 [0 to 10] | 4.8 [1 to 9]
  Pruritis NRS Score at Week 24: number analyzed (Participants) | 40 | 40 | 41 | 42 | 30
  Pruritis NRS Score at Week 24 | 4.0 [0 to 9] | 3.2 [0 to 10] | 2.2 [0 to 8] | 3.6 [0 to 9] | 4.3 [0 to 9]
  Pruritis NRS Score at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 27
  Pruritis NRS Score at Week 26 | 3.7 [0 to 9] | 3.0 [0 to 10] | 2.0 [0 to 9] | 3.3 [0 to 9] | 4.1 [0 to 9]
  Pruritis NRS Score at Week 28: number analyzed (Participants) | 36 | 38 | 38 | 40 | 26
  Pruritis NRS Score at Week 28 | 3.7 [0 to 10] | 3.1 [0 to 10] | 1.8 [0 to 9] | 3.1 [0 to 8] | 3.5 [0 to 8]
  Pruritis NRS Score at Week 30: number analyzed (Participants) | 34 | 38 | 38 | 40 | 25
  Pruritis NRS Score at Week 30 | 3.3 [0 to 9] | 2.5 [0 to 10] | 2.1 [0 to 9] | 2.9 [0 to 9] | 3.5 [0 to 9]
  Pruritis NRS Score at Week 32: number analyzed (Participants) | 33 | 37 | 37 | 40 | 24
  Pruritis NRS Score at Week 32 | 3.2 [0 to 9] | 2.7 [0 to 10] | 2.0 [0 to 9] | 2.7 [0 to 7] | 2.9 [0 to 8]
  Pruritis NRS Score at Week 34: number analyzed (Participants) | 33 | 37 | 36 | 37 | 24
  Pruritis NRS Score at Week 34 | 3.1 [0 to 9] | 2.8 [0 to 10] | 1.9 [0 to 7] | 3.0 [0 to 8] | 2.7 [0 to 8]
  Pruritis NRS Score at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 38 | 25
  Pruritis NRS Score at Week 36 | 3.1 [0 to 8] | 2.5 [0 to 10] | 1.8 [0 to 8] | 2.8 [0 to 8] | 2.6 [0 to 9]
  Pruritis NRS Score at Week 40: number analyzed (Participants) | 26 | 34 | 30 | 30 | 22
  Pruritis NRS Score at Week 40 | 2.8 [0 to 8] | 2.9 [0 to 10] | 2.1 [0 to 10] | 2.8 [0 to 8] | 2.4 [0 to 7]
  Pruritis NRS Score at Week 44: number analyzed (Participants) | 25 | 35 | 29 | 30 | 19
  Pruritis NRS Score at Week 44 | 2.9 [0 to 7] | 2.4 [0 to 10] | 1.6 [0 to 6] | 2.3 [0 to 8] | 1.6 [0 to 5]
  Pruritis NRS Score at Week 48: number analyzed (Participants) | 22 | 32 | 28 | 26 | 17
  Pruritis NRS Score at Week 48 | 3.2 [0 to 9] | 2.2 [0 to 10] | 1.7 [0 to 7] | 2.2 [0 to 6] | 1.8 [0 to 9]
  Pruritis NRS Score at Week 52: number analyzed (Participants) | 18 | 32 | 23 | 24 | 17
  Pruritis NRS Score at Week 52 | 2.8 [0 to 9] | 2.0 [0 to 10] | 1.9 [0 to 10] | 2.9 [0 to 10] | 1.4 [0 to 4]
  Pruritis NRS Score at Week 56: number analyzed (Participants) | 19 | 28 | 18 | 20 | 16
  Pruritis NRS Score at Week 56 | 2.8 [0 to 9] | 2.3 [0 to 10] | 1.9 [0 to 10] | 2.4 [0 to 10] | 1.3 [0 to 3]

21. Secondary Outcome: Percent Change From Baseline in Pruritus Numerical Rating Scale (NRS) Score at Each Time Point
Description: as for outcome 8
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change
  Pruritis NRS Score % Change at Week 1: number analyzed (Participants) | 50 | 52 | 51 | 54 | 54
  Pruritis NRS Score % Change at Week 1 | -2.9 [-60 to 167] | 2.5 [-56 to 250] | -3.4 [-88 to 100] | -12.2 [-50 to 33] | 2.6 [-67 to 300]
  Pruritis NRS Score % Change at Week 2: number analyzed (Participants) | 46 | 51 | 48 | 53 | 50
  Pruritis NRS Score % Change at Week 2 | -12.2 [-63 to 67] | -1.7 [-50 to 200] | -11.9 [-78 to 50] | -11.8 [-89 to 43] | 12.9 [-75 to 300]
  Pruritis NRS Score % Change at Week 4: number analyzed (Participants) | 46 | 49 | 46 | 52 | 44
  Pruritis NRS Score % Change at Week 4 | -16.8 [-80 to 80] | -8.3 [-80 to 250] | -18.8 [-100 to 133] | -17.3 [-89 to 43] | 14.0 [-63 to 350]
  Pruritis NRS Score % Change at Week 6: number analyzed (Participants) | 42 | 48 | 42 | 51 | 41
  Pruritis NRS Score % Change at Week 6 | -22.1 [-90 to 80] | -26.0 [-100 to 75] | -32.5 [-100 to 25] | -26.0 [-100 to 100] | 5.2 [-71 to 300]
  Pruritis NRS Score % Change at Week 8: number analyzed (Participants) | 42 | 45 | 42 | 50 | 40
  Pruritis NRS Score % Change at Week 8 | -28.1 [-90 to 60] | -25.5 [-100 to 200] | -37.3 [-100 to 50] | -31.0 [-89 to 33] | -8.8 [-88 to 200]
  Pruritis NRS Score % Change at Week 10: number analyzed (Participants) | 43 | 44 | 43 | 48 | 39
  Pruritis NRS Score % Change at Week 10 | -37.0 [-90 to 20] | -36.9 [-100 to 75] | -43.5 [-100 to 50] | -32.1 [-88 to 50] | -14.3 [-89 to 200]
  Pruritis NRS Score % Change at Week 12: number analyzed (Participants) | 43 | 45 | 42 | 48 | 36
  Pruritis NRS Score % Change at Week 12 | -37.9 [-100 to 29] | -37.9 [-100 to 250] | -49.0 [-100 to 33] | -36.0 [-90 to 40] | -16.0 [-89 to 100]
  Pruritis NRS Score % Change at Week 14: number analyzed (Participants) | 42 | 42 | 42 | 48 | 34
  Pruritis NRS Score % Change at Week 14 | -43.9 [-90 to 0] | -45.1 [-100 to 100] | -52.7 [-100 to 50] | -36.0 [-90 to 100] | -13.5 [-88 to 200]
  Pruritis NRS Score % Change at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  Pruritis NRS Score % Change at Week 15 | -41.7 [-90 to 29] | -43.6 [-100 to 150] | -57.8 [-100 to 25] | -42.6 [-90 to 20] | -16.3 [-89 to 300]
  Pruritis NRS Score % Change at Week 16: number analyzed (Participants) | 41 | 44 | 43 | 46 | 36
  Pruritis NRS Score % Change at Week 16 | -39.9 [-90 to 29] | -44.1 [-100 to 200] | -57.4 [-100 to 50] | -45.7 [-100 to 20] | -20.4 [-100 to 200]
  Pruritis NRS Score % Change at Week 18: number analyzed (Participants) | 41 | 43 | 40 | 46 | 33
  Pruritis NRS Score % Change at Week 18 | -45.8 [-89 to 13] | -44.5 [-100 to 250] | -52.1 [-100 to 25] | -42.9 [-100 to 100] | -29.3 [-100 to 60]
  Pruritis NRS Score % Change at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  Pruritis NRS Score % Change at Week 20 | -46.6 [-90 to 50] | -49.2 [-100 to 250] | -56.5 [-100 to 50] | -49.7 [-100 to 33] | -25.1 [-100 to 200]
  Pruritis NRS Score % Change at Week 22: number analyzed (Participants) | 39 | 40 | 42 | 45 | 31
  Pruritis NRS Score % Change at Week 22 | -48.0 [-100 to 13] | -52.1 [-100 to 250] | -66.2 [-100 to 25] | -53.6 [-100 to 11] | -20.9 [-90 to 300]
  Pruritis NRS Score % Change at Week 24: number analyzed (Participants) | 40 | 40 | 41 | 42 | 30
  Pruritis NRS Score % Change at Week 24 | -48.9 [-100 to 14] | -53.3 [-100 to 75] | -66.7 [-100 to 0] | -51.4 [-100 to 13] | -33.7 [-100 to 100]
  Pruritis NRS Score % Change at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 27
  Pruritis NRS Score % Change at Week 26 | -52.4 [-100 to 13] | -52.2 [-100 to 200] | -71.2 [-100 to 0] | -54.0 [-100 to 30] | -39.3 [-100 to 40]
  Pruritis NRS Score % Change at Week 28: number analyzed (Participants) | 36 | 38 | 38 | 40 | 26
  Pruritis NRS Score % Change at Week 28 | -50.3 [-100 to 40] | -56.2 [-100 to 11] | -73.7 [-100 to 25] | -57.1 [-100 to 0] | -45.4 [-100 to 20]
  Pruritis NRS Score % Change at Week 30: number analyzed (Participants) | 34 | 38 | 38 | 40 | 25
  Pruritis NRS Score % Change at Week 30 | -56.1 [-100 to 14] | -64.3 [-100 to 11] | -69.4 [-100 to 75] | -60.0 [-100 to 20] | -48.4 [-100 to 80]
  Pruritis NRS Score % Change at Week 32: number analyzed (Participants) | 33 | 37 | 37 | 40 | 24
  Pruritis NRS Score % Change at Week 32 | -58.3 [-100 to 13] | -61.4 [-100 to 11] | -70.5 [-100 to 25] | -60.9 [-100 to 20] | -63.6 [-100 to 0]
  Pruritis NRS Score % Change at Week 34: number analyzed (Participants) | 33 | 37 | 36 | 37 | 24
  Pruritis NRS Score % Change at Week 34 | -60.9 [-100 to 13] | -58.1 [-100 to 50] | -72.8 [-100 to 25] | -57.5 [-100 to 40] | -63.1 [-100 to 40]
  Pruritis NRS Score % Change at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 38 | 25
  Pruritis NRS Score % Change at Week 36 | -59.7 [-100 to 0] | -60.9 [-100 to 150] | -72.3 [-100 to 25] | -60.5 [-100 to 60] | -64.0 [-100 to 13]
  Pruritis NRS Score % Change at Week 40: number analyzed (Participants) | 26 | 34 | 30 | 30 | 22
  Pruritis NRS Score % Change at Week 40 | -61.7 [-100 to 0] | -52.8 [-100 to 250] | -70.2 [-100 to 25] | -60.7 [-100 to 0] | -67.0 [-100 to 0]
  Pruritis NRS Score % Change at Week 44: number analyzed (Participants) | 25 | 35 | 29 | 30 | 19
  Pruritis NRS Score % Change at Week 44 | -59.2 [-100 to 0] | -70.6 [-100 to 11] | -77.1 [-100 to -25] | -68.4 [-100 to 0] | -75.2 [-100 to -29]
  Pruritis NRS Score % Change at Week 48: number analyzed (Participants) | 22 | 32 | 28 | 26 | 17
  Pruritis NRS Score % Change at Week 48 | -56.7 [-100 to -10] | -69.3 [-100 to 11] | -74.0 [-100 to 0] | -68.3 [-100 to 0] | -69.7 [-100 to 80]
  Pruritis NRS Score % Change at Week 52: number analyzed (Participants) | 18 | 32 | 23 | 24 | 17
  Pruritis NRS Score % Change at Week 52 | -57.1 [-100 to 50] | -70.1 [-100 to 50] | -72.9 [-100 to 43] | -60.3 [-100 to 11] | -80.3 [-100 to 33]
  Pruritis NRS Score % Change at Week 56: number analyzed (Participants) | 19 | 28 | 18 | 20 | 16
  Pruritis NRS Score % Change at Week 56 | -60.2 [-100 to 0] | -67.2 [-100 to 14] | -75.7 [-100 to 0] | -65.6 [-100 to 11] | -82.1 [-100 to -50]

22. Secondary Outcome: Sleep Disturbance Numerical Rating Scale (NRS) Score at Each Time Point
Description: as for outcome 10
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale
  Sleep Disturbance NRS Score at Baseline | 5.9 [0 to 10] | 5.5 [0 to 10] | 5.0 [0 to 10] | 5.9 [0 to 10] | 5.0 [0 to 10]
  Sleep Disturbance NRS Score at Week 1: number analyzed (Participants) | 50 | 52 | 51 | 54 | 54
  Sleep Disturbance NRS Score at Week 1 | 6.0 [1 to 10] | 5.4 [0 to 10] | 5.2 [0 to 10] | 5.1 [0 to 10] | 5.1 [0 to 10]
  Sleep Disturbance NRS Score at Week 2: number analyzed (Participants) | 46 | 51 | 48 | 53 | 50
  Sleep Disturbance NRS Score at Week 2 | 5.3 [1 to 10] | 5.1 [0 to 10] | 4.7 [0 to 10] | 5.5 [0 to 10] | 5.6 [0 to 10]
  Sleep Disturbance NRS Score at Week 4: number analyzed (Participants) | 46 | 49 | 46 | 52 | 44
  Sleep Disturbance NRS Score at Week 4 | 5.5 [0 to 10] | 4.7 [0 to 10] | 4.3 [0 to 10] | 5.0 [0 to 10] | 5.6 [0 to 10]
  Sleep Disturbance NRS Score at Week 6: number analyzed (Participants) | 42 | 48 | 42 | 51 | 41
  Sleep Disturbance NRS Score at Week 6 | 5.3 [0 to 10] | 3.8 [0 to 10] | 3.2 [0 to 9] | 4.3 [0 to 9] | 5.0 [0 to 9]
  Sleep Disturbance NRS Score at Week 8: number analyzed (Participants) | 42 | 45 | 42 | 50 | 40
  Sleep Disturbance NRS Score at Week 8 | 4.5 [0 to 10] | 3.5 [0 to 10] | 3.0 [0 to 9] | 4.2 [0 to 10] | 4.8 [0 to 10]
  Sleep Disturbance NRS Score at Week 10: number analyzed (Participants) | 43 | 44 | 43 | 48 | 39
  Sleep Disturbance NRS Score at Week 10 | 3.9 [0 to 9] | 3.1 [0 to 10] | 2.5 [0 to 8] | 3.9 [0 to 9] | 4.6 [0 to 10]
  Sleep Disturbance NRS Score at Week 12: number analyzed (Participants) | 43 | 45 | 42 | 48 | 36
  Sleep Disturbance NRS Score at Week 12 | 3.5 [0 to 10] | 3.2 [0 to 9] | 2.1 [0 to 9] | 3.6 [0 to 10] | 4.4 [0 to 9]
  Sleep Disturbance NRS Score at Week 14: number analyzed (Participants) | 42 | 42 | 42 | 48 | 34
  Sleep Disturbance NRS Score at Week 14 | 3.8 [0 to 9] | 2.5 [0 to 9] | 2.5 [0 to 8] | 3.3 [0 to 10] | 4.7 [0 to 10]
  Sleep Disturbance NRS Score at Week 15: number analyzed (Participants) | 40 | 43 | 41 | 48 | 37
  Sleep Disturbance NRS Score at Week 15 | 3.4 [0 to 9] | 2.7 [0 to 9] | 1.9 [0 to 8] | 3.0 [0 to 7] | 4.6 [0 to 9]
  Sleep Disturbance NRS Score at Week 16: number analyzed (Participants) | 41 | 44 | 43 | 47 | 36
  Sleep Disturbance NRS Score at Week 16 | 3.5 [0 to 10] | 2.7 [0 to 8] | 1.8 [0 to 7] | 2.9 [0 to 8] | 4.2 [0 to 10]
  Sleep Disturbance NRS Score at Week 18: number analyzed (Participants) | 41 | 43 | 40 | 46 | 33
  Sleep Disturbance NRS Score at Week 18 | 3.6 [0 to 9] | 2.3 [0 to 9] | 1.6 [0 to 6] | 3.2 [0 to 10] | 4.2 [0 to 9]
  Sleep Disturbance NRS Score at Week 20: number analyzed (Participants) | 41 | 41 | 39 | 45 | 30
  Sleep Disturbance NRS Score at Week 20 | 3.1 [0 to 10] | 2.1 [0 to 8] | 1.6 [0 to 7] | 2.9 [0 to 10] | 4.0 [0 to 9]
  Sleep Disturbance NRS Score at Week 22: number analyzed (Participants) | 39 | 40 | 42 | 45 | 31
  Sleep Disturbance NRS Score at Week 22 | 3.1 [0 to 9] | 2.3 [0 to 9] | 1.3 [0 to 6] | 2.7 [0 to 10] | 3.8 [0 to 9]
  Sleep Disturbance NRS Score at Week 24: number analyzed (Participants) | 40 | 40 | 41 | 42 | 30
  Sleep Disturbance NRS Score at Week 24 | 2.9 [0 to 9] | 2.1 [0 to 8] | 1.5 [0 to 9] | 2.7 [0 to 8] | 3.5 [0 to 9]
  Sleep Disturbance NRS Score at Week 26: number analyzed (Participants) | 38 | 38 | 39 | 43 | 27
  Sleep Disturbance NRS Score at Week 26 | 3.1 [0 to 9] | 1.7 [0 to 7] | 1.2 [0 to 5] | 2.4 [0 to 8] | 3.2 [0 to 9]
  Sleep Disturbance NRS Score at Week 28: number analyzed (Participants) | 36 | 38 | 38 | 40 | 26
  Sleep Disturbance NRS Score at Week 28 | 3.1 [0 to 10] | 1.6 [0 to 7] | 1.1 [0 to 7] | 2.3 [0 to 8] | 2.7 [0 to 8]
  Sleep Disturbance NRS Score at Week 30: number analyzed (Participants) | 34 | 38 | 38 | 40 | 25
  Sleep Disturbance NRS Score at Week 30 | 2.5 [0 to 9] | 1.4 [0 to 7] | 1.1 [0 to 6] | 1.9 [0 to 9] | 2.6 [0 to 9]
  Sleep Disturbance NRS Score at Week 32: number analyzed (Participants) | 33 | 38 | 37 | 40 | 24
  Sleep Disturbance NRS Score at Week 32 | 2.3 [0 to 9] | 1.9 [0 to 8] | 1.2 [0 to 5] | 1.9 [0 to 8] | 2.4 [0 to 8]
  Sleep Disturbance NRS Score at Week 34: number analyzed (Participants) | 33 | 37 | 36 | 37 | 24
  Sleep Disturbance NRS Score at Week 34 | 2.3 [0 to 9] | 1.5 [0 to 8] | 0.9 [0 to 6] | 2.1 [0 to 7] | 2.1 [0 to 8]
  Sleep Disturbance NRS Score at Week 36: number analyzed (Participants) | 34 | 37 | 36 | 38 | 25
  Sleep Disturbance NRS Score at Week 36 | 2.0 [0 to 9] | 1.6 [0 to 8] | 0.9 [0 to 6] | 2.1 [0 to 8] | 2.0 [0 to 9]
  Sleep Disturbance NRS Score at Week 40: number analyzed (Participants) | 27 | 34 | 30 | 30 | 22
  Sleep Disturbance NRS Score at Week 40 | 1.5 [0 to 8] | 1.5 [0 to 7] | 0.8 [0 to 4] | 1.9 [0 to 7] | 2.0 [0 to 8]
  Sleep Disturbance NRS Score at Week 44: number analyzed (Participants) | 25 | 35 | 29 | 30 | 19
  Sleep Disturbance NRS Score at Week 44 | 1.9 [0 to 7] | 1.4 [0 to 8] | 0.6 [0 to 4] | 1.4 [0 to 8] | 1.1 [0 to 4]
  Sleep Disturbance NRS Score at Week 48: number analyzed (Participants) | 22 | 32 | 28 | 26 | 17
  Sleep Disturbance NRS Score at Week 48 | 2.1 [0 to 9] | 1.2 [0 to 8] | 0.6 [0 to 4] | 1.3 [0 to 5] | 0.9 [0 to 2]
  Sleep Disturbance NRS Score at Week 52: number analyzed (Participants) | 18 | 32 | 23 | 24 | 17
  Sleep Disturbance NRS Score at Week 52 | 1.6 [0 to 7] | 0.8 [0 to 8] | 1.3 [0 to 9] | 1.9 [0 to 6] | 1.2 [0 to 3]
  Sleep Disturbance NRS Score at Week 56: number analyzed (Participants) | 19 | 28 | 18 | 20 | 16
  Sleep Disturbance NRS Score at Week 56 | 2.1 [0 to 9] | 1.1 [0 to 8] | 1.1 [0 to 9] | 1.5 [0 to 8] | 0.9 [0 to 2]

23. Secondary Outcome: Percent Change From Baseline in Sleep Disturbance Numerical Rating Scale (NRS) Score at Each Time Point
Description: as for outcome 10
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: percentage of score change
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
percentage of score change
  Sleep Disturbance NRS Score % Change at Week 1: number analyzed (Participants) | 49 | 47 | 46 | 51 | 51
  Sleep Disturbance NRS Score % Change at Week 1 | 6.6 [-83 to 300] | 14.2 [-100 to 500] | 29.8 [-100 to 400] | -15.7 [-100 to 80] | 51.3 [-100 to 700]
  Sleep Disturbance NRS Score % Change at Week 2: number analyzed (Participants) | 45 | 46 | 43 | 50 | 47
  Sleep Disturbance NRS Score % Change at Week 2 | -0.7 [-90 to 350] | 12.6 [-100 to 600] | 12.0 [-100 to 350] | -6.7 [-100 to 167] | 60.3 [-100 to 700]
  Sleep Disturbance NRS Score % Change at Week 4: number analyzed (Participants) | 45 | 44 | 41 | 49 | 41
  Sleep Disturbance NRS Score % Change at Week 4 | 4.9 [-100 to 400] | 12.1 [-100 to 500] | 11.9 [-100 to 600] | -11.2 [-100 to 167] | 49.6 [-100 to 600]
  Sleep Disturbance NRS Score % Change at Week 6: number analyzed (Participants) | 41 | 43 | 37 | 48 | 38
  Sleep Disturbance NRS Score % Change at Week 6 | 6.2 [-100 to 400] | -7.1 [-100 to 500] | -18.3 [-100 to 400] | -25.5 [-100 to 167] | 33.6 [-100 to 500]
  Sleep Disturbance NRS Score % Change at Week 8: number analyzed (Participants) | 41 | 40 | 37 | 47 | 37
  Sleep Disturbance NRS Score % Change at Week 8 | -11.7 [-100 to 300] | -10.8 [-100 to 400] | -27.3 [-100 to 400] | -31.8 [-100 to 43] | 13.5 [-100 to 500]
  Sleep Disturbance NRS Score % Change at Week 10: number analyzed (Participants) | 42 | 39 | 38 | 45 | 37
  Sleep Disturbance NRS Score % Change at Week 10 | -29.8 [-100 to 300] | -31.9 [-100 to 200] | -41.3 [-100 to 200] | -36.1 [-100 to 60] | 11.7 [-100 to 500]
  Sleep Disturbance NRS Score % Change at Week 12: number analyzed (Participants) | 42 | 40 | 37 | 45 | 34
  Sleep Disturbance NRS Score % Change at Week 12 | -37.1 [-100 to 200] | -13.4 [-100 to 500] | -54.8 [-100 to 17] | -38.9 [-100 to 33] | 4.5 [-100 to 500]
  Sleep Disturbance NRS Score % Change at Week 14: number analyzed (Participants) | 41 | 38 | 37 | 45 | 32
  Sleep Disturbance NRS Score % Change at Week 14 | -34.5 [-100 to 200] | -38.4 [-100 to 400] | -49.6 [-100 to 50] | -44.0 [-100 to 40] | 14.5 [-100 to 600]
  Sleep Disturbance NRS Score % Change at Week 15: number analyzed (Participants) | 39 | 38 | 36 | 45 | 35
  Sleep Disturbance NRS Score % Change at Week 15 | -41.9 [-100 to 100] | -28.1 [-100 to 300] | -60.9 [-100 to 100] | -46.6 [-100 to 25] | 13.7 [-100 to 500]
  Sleep Disturbance NRS Score % Change at Week 16: number analyzed (Participants) | 40 | 39 | 38 | 44 | 34
  Sleep Disturbance NRS Score % Change at Week 16 | -38.4 [-100 to 100] | -10.9 [-100 to 600] | -63.4 [-100 to 67] | -48.5 [-100 to 50] | 0.7 [-100 to 600]
  Sleep Disturbance NRS Score % Change at Week 18: number analyzed (Participants) | 40 | 39 | 35 | 43 | 32
  Sleep Disturbance NRS Score % Change at Week 18 | -42.2 [-100 to 50] | -48.7 [-100 to 300] | -66.9 [-100 to 25] | -38.9 [-100 to 300] | 8.1 [-100 to 700]
  Sleep Disturbance NRS Score % Change at Week 20: number analyzed (Participants) | 40 | 37 | 34 | 42 | 28
  Sleep Disturbance NRS Score % Change at Week 20 | -44.4 [-100 to 100] | -48.4 [-100 to 500] | -72.3 [-100 to 25] | -50.0 [-100 to 50] | 9.1 [-100 to 800]
  Sleep Disturbance NRS Score % Change at Week 22: number analyzed (Participants) | 38 | 36 | 37 | 42 | 29
  Sleep Disturbance NRS Score % Change at Week 22 | -45.0 [-100 to 200] | -45.1 [-100 to 500] | -75.1 [-100 to 25] | -56.1 [-100 to 29] | -2.3 [-100 to 700]
  Sleep Disturbance NRS Score % Change at Week 24: number analyzed (Participants) | 39 | 37 | 37 | 39 | 28
  Sleep Disturbance NRS Score % Change at Week 24 | -53.1 [-100 to 50] | -53.3 [-100 to 200] | -67.3 [-100 to 200] | -52.5 [-100 to 60] | -5.5 [-100 to 600]
  Sleep Disturbance NRS Score % Change at Week 26: number analyzed (Participants) | 38 | 35 | 35 | 40 | 25
  Sleep Disturbance NRS Score % Change at Week 26 | -46.5 [-100 to 100] | -55.5 [-100 to 300] | -75.5 [-100 to 0] | -57.1 [-100 to 60] | -39.4 [-100 to 80]
  Sleep Disturbance NRS Score % Change at Week 28: number analyzed (Participants) | 35 | 35 | 34 | 37 | 24
  Sleep Disturbance NRS Score % Change at Week 28 | -48.7 [-100 to 100] | -54.4 [-100 to 200] | -80.4 [-100 to 50] | -58.8 [-100 to 33] | -38.9 [-100 to 60]
  Sleep Disturbance NRS Score % Change at Week 30: number analyzed (Participants) | 33 | 35 | 34 | 37 | 23
  Sleep Disturbance NRS Score % Change at Week 30 | -58.1 [-100 to 29] | -63.3 [-100 to 300] | -77.4 [-100 to 67] | -67.1 [-100 to 40] | -45.6 [-100 to 80]
  Sleep Disturbance NRS Score % Change at Week 32: number analyzed (Participants) | 32 | 35 | 33 | 37 | 22
  Sleep Disturbance NRS Score % Change at Week 32 | -60.0 [-100 to 0] | -45.6 [-100 to 700] | -78.0 [-100 to 25] | -65.8 [-100 to 0] | -55.3 [-100 to 40]
  Sleep Disturbance NRS Score % Change at Week 34: number analyzed (Participants) | 32 | 34 | 32 | 34 | 22
  Sleep Disturbance NRS Score % Change at Week 34 | -61.1 [-100 to 0] | -66.0 [-100 to 100] | -82.5 [-100 to 0] | -64.8 [-100 to 20] | -51.7 [-100 to 33]
  Sleep Disturbance NRS Score % Change at Week 36: number analyzed (Participants) | 33 | 34 | 32 | 35 | 23
  Sleep Disturbance NRS Score % Change at Week 36 | -64.9 [-100 to 17] | -45.1 [-100 to 700] | -81.9 [-100 to -25] | -64.7 [-100 to 20] | -56.2 [-100 to 20]
  Sleep Disturbance NRS Score % Change at Week 40: number analyzed (Participants) | 26 | 31 | 26 | 28 | 20
  Sleep Disturbance NRS Score % Change at Week 40 | -71.6 [-100 to 0] | -50.7 [-100 to 400] | -81.0 [-100 to 0] | -67.8 [-100 to 0] | -57.2 [-100 to 60]
  Sleep Disturbance NRS Score % Change at Week 44: number analyzed (Participants) | 25 | 32 | 25 | 28 | 17
  Sleep Disturbance NRS Score % Change at Week 44 | -65.7 [-100 to 25] | -71.4 [-100 to 100] | -88.5 [-100 to 0] | -79.6 [-100 to -14] | -65.3 [-100 to 0]
  Sleep Disturbance NRS Score % Change at Week 48: number analyzed (Participants) | 22 | 29 | 24 | 24 | 15
  Sleep Disturbance NRS Score % Change at Week 48 | -60.0 [-100 to 33] | -70.2 [-100 to 100] | -84.9 [-100 to 33] | -78.9 [-100 to -25] | -74.4 [-100 to 0]
  Sleep Disturbance NRS Score % Change at Week 52: number analyzed (Participants) | 18 | 29 | 20 | 22 | 15
  Sleep Disturbance NRS Score % Change at Week 52 | -73.2 [-100 to 17] | -87.0 [-100 to 14] | -61.9 [-100 to 200] | -71.1 [-100 to -14] | -69.3 [-100 to 0]
  Sleep Disturbance NRS Score % Change at Week 56: number analyzed (Participants) | 19 | 25 | 16 | 18 | 14
  Sleep Disturbance NRS Score % Change at Week 56 | -65.9 [-100 to 50] | -69.7 [-100 to 200] | -82.2 [-100 to 0] | -75.9 [-100 to 0] | -71.3 [-100 to 0]

24. Secondary Outcome: Dermatology Life Quality Index (DLQI) at Each Time Point
Description: as for outcome 12
Time Frame: 56 Weeks
Population: as for outcome 13
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
Number analyzed (Participants) | 52 | 52 | 52 | 54 | 57
score on a scale
  DLQI Score at Baseline: number analyzed (Participants) | 48 | 45 | 47 | 48 | 52
  DLQI Score at Baseline | 13.4 [2 to 30] | 12.6 [1 to 29] | 12.0 [1 to 27] | 13.8 [1 to 27] | 11.9 [2 to 30]
  DLQI Score at Week 1: number analyzed (Participants) | 47 | 43 | 45 | 46 | 48
  DLQI Score at Week 1 | 14.1 [2 to 29] | 12.8 [1 to 29] | 11.2 [1 to 27] | 12.7 [1 to 27] | 12.2 [1 to 30]
  DLQI Score at Week 2: number analyzed (Participants) | 42 | 42 | 42 | 45 | 41
  DLQI Score at Week 2 | 12.6 [1 to 30] | 12.6 [0 to 30] | 10.7 [1 to 28] | 12.7 [3 to 29] | 12.3 [2 to 27]
  DLQI Score at Week 4: number analyzed (Participants) | 42 | 42 | 40 | 44 | 37
  DLQI Score at Week 4 | 12.5 [0 to 29] | 12.7 [0 to 29] | 10.2 [1 to 28] | 11.2 [1 to 28] | 13.3 [1 to 30]
  DLQI Score at Week 6: number analyzed (Participants) | 40 | 42 | 37 | 42 | 35
  DLQI Score at Week 6 | 11.3 [0 to 29] | 10.2 [0 to 27] | 7.1 [1 to 20] | 9.6 [0 to 29] | 10.7 [1 to 30]
  DLQI Score at Week 8: number analyzed (Participants) | 36 | 41 | 38 | 44 | 34
  DLQI Score at Week 8 | 9.7 [0 to 26] | 8.9 [0 to 25] | 7.1 [0 to 17] | 9.0 [1 to 29] | 11.4 [1 to 29]
  DLQI Score at Week 10: number analyzed (Participants) | 38 | 39 | 35 | 42 | 31
  DLQI Score at Week 10 | 8.0 [0 to 27] | 8.0 [1 to 22] | 7.1 [1 to 21] | 8.3 [1 to 28] | 10.6 [1 to 26]
  DLQI Score at Week 12: number analyzed (Participants) | 38 | 38 | 35 | 42 | 31
  DLQI Score at Week 12 | 7.6 [0 to 26] | 7.2 [0 to 21] | 5.8 [0 to 19] | 7.8 [0 to 30] | 9.7 [0 to 24]
  DLQI Score at Week 14: number analyzed (Participants) | 39 | 39 | 35 | 43 | 28
  DLQI Score at Week 14 | 7.4 [0 to 21] | 6.9 [0 to 19] | 5.1 [0 to 16] | 7.2 [1 to 23] | 10.1 [1 to 28]
  DLQI Score at Week 15: number analyzed (Participants) | 36 | 36 | 35 | 42 | 31
  DLQI Score at Week 15 | 7.5 [1 to 25] | 6.2 [0 to 17] | 4.4 [0 to 16] | 5.9 [0 to 18] | 10.3 [0 to 28]
  DLQI Score at Week 16: number analyzed (Participants) | 36 | 39 | 37 | 41 | 32
  DLQI Score at Week 16 | 7.6 [0 to 21] | 6.1 [0 to 19] | 4.7 [0 to 14] | 6.7 [0 to 20] | 9.8 [0 to 27]
  DLQI Score at Week 18: number analyzed (Participants) | 36 | 39 | 34 | 40 | 30
  DLQI Score at Week 18 | 6.7 [0 to 24] | 6.7 [0 to 21] | 4.9 [0 to 16] | 6.6 [0 to 23] | 9.5 [0 to 29]
  DLQI Score at Week 20: number analyzed (Participants) | 35 | 36 | 33 | 40 | 26
  DLQI Score at Week 20 | 6.7 [0 to 27] | 6.2 [0 to 23] | 5.0 [0 to 17] | 5.6 [0 to 20] | 8.8 [0 to 23]
  DLQI Score at Week 22: number analyzed (Participants) | 35 | 35 | 38 | 40 | 26
  DLQI Score at Week 22 | 6.3 [0 to 25] | 5.8 [0 to 19] | 4.3 [0 to 19] | 5.3 [0 to 21] | 8.6 [0 to 25]
  DLQI Score at Week 24: number analyzed (Participants) | 35 | 35 | 36 | 37 | 25
  DLQI Score at Week 24 | 6.8 [0 to 25] | 5.4 [0 to 20] | 4.3 [0 to 17] | 5.1 [0 to 14] | 8.0 [0 to 27]
  DLQI Score at Week 26: number analyzed (Participants) | 33 | 36 | 33 | 40 | 22
  DLQI Score at Week 26 | 6.7 [0 to 28] | 5.2 [0 to 17] | 3.7 [0 to 14] | 5.2 [0 to 16] | 7.5 [0 to 27]
  DLQI Score at Week 28: number analyzed (Participants) | 32 | 36 | 32 | 35 | 22
  DLQI Score at Week 28 | 6.8 [0 to 26] | 5.0 [0 to 13] | 3.3 [0 to 10] | 4.4 [0 to 14] | 6.6 [1 to 26]
  DLQI Score at Week 30: number analyzed (Participants) | 31 | 36 | 33 | 37 | 23
  DLQI Score at Week 30 | 6.0 [0 to 24] | 4.4 [0 to 13] | 3.9 [0 to 18] | 4.0 [0 to 18] | 6.9 [0 to 25]
  DLQI Score at Week 32: number analyzed (Participants) | 28 | 35 | 33 | 38 | 22
  DLQI Score at Week 32 | 5.8 [0 to 30] | 5.3 [0 to 16] | 3.6 [0 to 16] | 3.5 [0 to 11] | 6.1 [0 to 26]
  DLQI Score at Week 34: number analyzed (Participants) | 29 | 34 | 31 | 35 | 22
  DLQI Score at Week 34 | 5.3 [0 to 30] | 5.3 [0 to 20] | 2.9 [0 to 15] | 3.7 [0 to 11] | 4.9 [0 to 25]
  DLQI Score at Week 36: number analyzed (Participants) | 30 | 35 | 31 | 36 | 21
  DLQI Score at Week 36 | 5.1 [0 to 24] | 4.5 [0 to 13] | 2.9 [0 to 10] | 3.6 [0 to 18] | 4.4 [0 to 25]
  DLQI Score at Week 40: number analyzed (Participants) | 24 | 33 | 27 | 27 | 20
  DLQI Score at Week 40 | 3.7 [0 to 20] | 4.8 [0 to 20] | 3.3 [0 to 11] | 3.7 [0 to 10] | 4.1 [0 to 24]
  DLQI Score at Week 44: number analyzed (Participants) | 21 | 33 | 27 | 27 | 17
  DLQI Score at Week 44 | 3.5 [0 to 16] | 3.7 [0 to 21] | 3.3 [0 to 10] | 3.3 [0 to 10] | 1.9 [0 to 24]
  DLQI Score at Week 48: number analyzed (Participants) | 19 | 31 | 25 | 24 | 14
  DLQI Score at Week 48 | 4.6 [0 to 19] | 3.1 [0 to 12] | 3.2 [0 to 10] | 2.9 [0 to 10] | 3.1 [0 to 17]
  DLQI Score at Week 52: number analyzed (Participants) | 15 | 31 | 23 | 23 | 14
  DLQI Score at Week 52 | 4.1 [0 to 27] | 3.1 [0 to 12] | 3.7 [0 to 23] | 3.8 [0 to 16] | 3.3 [0 to 19]
  DLQI Score at Week 56: number analyzed (Participants) | 17 | 27 | 16 | 19 | 13
  DLQI Score at Week 56 | 5.1 [0 to 15] | 3.4 [0 to 13] | 2.8 [0 to 8] | 4.7 [0 to 28] | 3.2 [0 to 22]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for reporting from the subject's written consent to participate in the study through the end of the study, up to 62 weeks (potential 6 week screening period up to Week 56).
Arm/Group | KHK4083 150 mg SC Q4W | KHK4083 600 mg SC Q4W | KHK4083 300 mg SC Q2W | KHK4083 600 mg SC Q2W | Placebo/KHK4083 600 mg
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/53 | 0/55 | 0/54 | 0/57
Serious Adverse Events (participants affected / at risk) | 4/54 | 1/53 | 4/55 | 1/54 | 2/57
Other Adverse Events (participants affected / at risk) | 47/54 | 50/53 | 48/55 | 51/54 | 46/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KHK4083 150 mg SC Q4W (N=54) | KHK4083 600 mg SC Q4W (N=53) | KHK4083 300 mg SC Q2W (N=55) | KHK4083 600 mg SC Q2W (N=54) | Placebo/KHK4083 600 mg (N=57)
Atopic cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestine ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KHK4083 150 mg SC Q4W (N=54) | KHK4083 600 mg SC Q4W (N=53) | KHK4083 300 mg SC Q2W (N=55) | KHK4083 600 mg SC Q2W (N=54) | Placebo/KHK4083 600 mg (N=57)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 3 (3) | 11 (18) | 4 (5) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (6) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (7) | 3 (3) | 2 (2) | 8 (8) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (10) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (3) | 1 (2) | 2 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 3 (3) | 7 (10) | 12 (14) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Injection site pain (General disorders) | 2 (4) | 3 (4) | 1 (13) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (5) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 9 (9) | 10 (11) | 11 (11) | 3 (3)
Influenza (Infections and infestations) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Kaposi's varicelliform eruption (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 13 (21) | 11 (16) | 12 (16) | 19 (25) | 13 (18)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 4 (6) | 4 (4) | 3 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Tinea pedis (Infections and infestations) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 4 (5) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (12) | 6 (9) | 6 (20) | 5 (6) | 5 (6)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 4 (6) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6) | 7 (8) | 3 (4) | 3 (3)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 19 (21) | 12 (12) | 18 (21) | 20 (22) | 24 (28)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03703102/Prot_SAP_000.pdf